CLINICAL TRIAL: NCT04889209
Title: A Phase 1/2 Study of Delayed Heterologous SARS-CoV-2 Vaccine Dosing (Boost) After Receipt of EUA Vaccines
Brief Title: Delayed Heterologous SARS-CoV-2 Vaccine Dosing (Boost) After Receipt of EUA Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-0012; 5UM1AI148684-02 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-05-17 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-07-08

CONDITIONS: COVID-19
Keywords: Heterologous Nonvariant Boost; SARS-COV-2; SARS-COV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Masking Description: study sites will administer product to which they have been assigned
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (18):
- Cohort 1 Group 10E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (boost dose). N = 50
  Interventions: Biological: mRNA-1273.211
- Cohort 1 Group 11E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (boost dose). N = 50
  Interventions: Biological: mRNA-1273.211
- Cohort 1 Group 12E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA- 1273 N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 13E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 14E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 15E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp for one or two doses stratified with two age ranges of 18-55 years (n= 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  Interventions: Biological: SARS-CoV-2 rS/M1
- Cohort 1 Group 16E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  Interventions: Biological: SARS-CoV-2 rS/M1
- Cohort 1 Group 17E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  Interventions: Biological: SARS-CoV-2 rS/M1
- Cohort 1 Group 1E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of 100-mcg dose of mRNA-1273 (boost dose). N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 2E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose). N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 3E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n ˜ 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose). N = 50
  Interventions: Biological: mRNA-1273
- Cohort 1 Group 4E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Interventions: Biological: Ad26.COV2.S
- Cohort 1 Group 5E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Interventions: Biological: Ad26.COV2.S
- Cohort 1 Group 6E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Interventions: Biological: Ad26.COV2.S
- Cohort 1 Group 7E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp stratified with two age ranges of 18-55 years (n=˜ 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose). N = 50
  Interventions: Biological: BNT162b2
- Cohort 1 Group 8E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose). N = 50
  Interventions: Biological: BNT162b2
- Cohort 1 Group 9E (Experimental): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose). N = 50
  Interventions: Biological: BNT162b2
- Cohort 2 (Experimental): A prospective design cohort with naïve to COVID-19 vaccine and infection participants of > / = 18 years of age to receive COVID-19 vaccine intramuscularly under Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at the 100mcg dose at a 28 days of interval) followed by a delayed vaccination (50 mcg mRNA-1273) after a minimum of 12 weeks. A second booster (fourth dose) will be administered intramuscular using Moderna mRNA-1273.222 at 50 mcg at a 4-12 month interval N=250
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.222

INTERVENTIONS:
Biological: Ad26.COV2.S — Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-ß-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
  Arms: Cohort 1 Group 4E; Cohort 1 Group 5E; Cohort 1 Group 6E
Biological: BNT162b2 — A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
  Arms: Cohort 1 Group 7E; Cohort 1 Group 8E; Cohort 1 Group 9E
Biological: mRNA-1273 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV). Doses are either 0.25 mL or 0.5 mL.
  Arms: Cohort 1 Group 12E; Cohort 1 Group 13E; Cohort 1 Group 14E; Cohort 1 Group 1E; Cohort 1 Group 2E; Cohort 1 Group 3E; Cohort 2
Biological: mRNA-1273.211 — Lipid nanoparticle (LNP) dispersion containing 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the B.1.351 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273. mRNA-1273.211 (0.2 mg/mL) will be administered in 0.5 mL doses (100 mcg/0.5 mL).
  Arms: Cohort 1 Group 10E; Cohort 1 Group 11E
Biological: mRNA-1273.222 — Formulated in the same way as the mRNA-1273 vaccine but contains 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273.
  Arms: Cohort 2
Biological: SARS-CoV-2 rS/M1 — SARS-CoV-2 rS Drug Substance containing the prototype Wuhan is formulated with saponin-based Matrix-M adjuvant in a buffer of 25 mM sodium phosphate (pH 7.2), 300 mM sodium chloride, and 0.01% (weight per volume [w/v]) polysorbate 80. NVX-Co-V2373 will be administered in 0.5 mL dose (5 mcg Prototype SARS-CoV-2 rS with 50 mcg Matrix-M adjuvant)
  Arms: Cohort 1 Group 15E; Cohort 1 Group 16E; Cohort 1 Group 17E

SUMMARY:
A phase 1/2, open-label clinical trial in individuals, 18 years of age and older, who are in good health, have no known history of Coronavirus Disease 2019 (COVID-19) or Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of a delayed (>/=12 weeks) vaccine boost on a range of Emergency Use Authorization (EUA)-dosed COVID-19 vaccines (mRNA-1273, and mRNA-1273.211 manufactured by ModernaTX, Inc.; BNT162b2 manufactured by Pfizer/BioNTech; or Ad26.COV2.S manufactured by Janssen Pharmaceuticals/Johnson & Johnson). This is an adaptive design and may add arms (and increase sample size) as vaccines are awarded EUA and/or variant lineage spike vaccines are manufactured or become available. Enrollment will occur at up to twelve domestic clinical research sites.

This study includes two cohorts. Cohort 1 will include approximately 880 individuals (50 subjects/group; Groups 1E-11E) greater than 18 years of age and older, stratified into two age strata (18-55 years and >/=56 years) who previously received COVID-19 vaccine at Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at the 100 mcg dose, two vaccinations of BNT162b2 at the 30 mcg dose, or one vaccination of Ad26.COV2.S at the 5x10^10 vp dose). Groups 15E-17E will enroll 60 subjects, split (approximately evenly) between age strata as able. Those subjects will be offered enrollment into this study >/=12 weeks after they received the last dose of their EUA vaccine. Subjects will receive a single open-label intramuscular (IM) injection of the designated delayed booster vaccine and will be followed through 12 months after vaccination: 1) Group 1E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp followed by a 100-mcg dose of mRNA-1273, Group 4E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 7E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp followed by a 30-mcg dose of BNT162b2, Group 10E - previously EUA-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp followed by a 100-mcg dose of mRNA-1273.211; Group 12E - previously EUA-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp followed by a 50-mcg dose of mRNA-1273; Group 15E - previously EUA-dosed vaccination with Janssen (two doses for Group 15E) - Ad26.COV2.S at 5x1010 vp followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV-2 rS vaccine with 50 mcg Matrix-M); 2) Group 2E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 100-mcg dose of mRNA-1273, Group 5E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 8E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 30-mcg dose of BNT162b2, Group 13E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 50-mcg dose of mRNA-1273; Group 16E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV2 rS vaccine with 50 mcg Matrix-M); 3) Group 3E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 100-mcg dose of mRNA-1273. Group 6E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 9E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 30-mcg dose of BNT162b2, Group 11E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 100-mcg dose of mRNA-1273.211. Group 14E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 50-mcg dose of mRNA-1273, Group 17E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV2 rS vaccine with 50 mcg Matrix-M).

A telephone visit will occur one week after each primary EUA vaccination and one week after the booster dose. In person follow-up visits will occur on 14 days following completion of EUA vaccinations and on days 14, and 28 days after the booster dose, as well as 3, 6, and 12 months post the booster vaccination. Additional pools of subjects can be included if needed as additional COVID-19 vaccines are awarded EUA.

The primary objectives of this study are 1) to evaluate the safety and reactogenicity of delayed heterologous or homologous vaccine doses after EUA dosed vaccines, and 2) to evaluate the breadth of the humoral immune responses of heterologous and homologous delayed boost regimens following EUA dosing.

DETAILED DESCRIPTION:
A phase 1/2, open-label clinical trial in individuals, 18 years of age and older, who are in good health, have no known history of Coronavirus Disease 2019 (COVID-19) or Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of a delayed (>/=12 weeks) vaccine boost on a range of Emergency Use Authorization (EUA)-dosed COVID-19 vaccines (mRNA-1273, and mRNA-1273.211 manufactured by ModernaTX, Inc.; BNT162b2 manufactured by Pfizer/BioNTech; or Ad26.COV2.S manufactured by Janssen Pharmaceuticals/Johnson & Johnson). This is an adaptive design and may add arms (and increase sample size) as vaccines are awarded EUA and/or variant lineage spike vaccines are manufactured or become available. Enrollment will occur at up to twelve domestic clinical research sites.

This study includes two cohorts. Cohort 1 will include approximately 880 individuals (50 subjects/group; Groups 1E-14E, and 60 subjects/group; Groups 15E-17E) greater than 18 years of age and older, stratified into two age strata (18-55 years and >/=56 years) who previously received COVID-19 vaccine at Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at the 100 mcg dose, two vaccinations of BNT162b2 at the 30 mcg dose, or one vaccination of Ad26.COV2.S at the 5x10^10 vp dose). Groups 15E-17E will enroll 60 subjects, split (approximately evenly) between age strata as able. Those subjects will be offered enrollment into this study >/=12 weeks after they received the last dose of their EUA vaccine. Subjects will receive a single open-label intramuscular (IM) injection of the designated delayed booster vaccine and will be followed through 12 months after vaccination: 1) Group 1E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp followed by a 100-mcg dose of mRNA-1273, Group 4E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 7E - previously EUA-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp followed by a 30-mcg dose of BNT162b2, Group 10E - previously EUA-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp followed by a 100-mcg dose of mRNA-1273.211; Group 12E - previously EUA-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp followed by a 50-mcg dose of mRNA-1273; Group 15E - previously EUA-dosed vaccination with Janssen (two doses for Group 15E) - Ad26.COV2.S at 5x1010 vp followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV-2 rS vaccine with 50 mcg Matrix-M); 2) Group 2E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 100-mcg dose of mRNA-1273, Group 5E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 8E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 30-mcg dose of BNT162b2, Group 13E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a 50-mcg dose of mRNA-1273; Group 16E - previously EUA-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV2 rS vaccine with 50 mcg Matrix-M); 3) Group 3E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 100-mcg dose of mRNA-1273. Group 6E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 5x10^10 vp dose of Ad26.COV2.S, Group 9E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 30-mcg dose of BNT162b2, Group 11E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 100-mcg dose of mRNA-1273.211. Group 14E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a 50-mcg dose of mRNA-1273, Group 17E - previously EUA-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses followed by a dose of NVX-CoV2373 (5 mcg Prototype SARS-CoV2 rS vaccine with 50 mcg Matrix-M).

A telephone visit will occur at Day 8 and in-person follow-up visits will occur on Days 15 and 29, as well as 3, 6, and 12 months after the vaccination. Cohort 2 will include approximately 250 participants per group aged >/=18 years of age who have not received a Coronavirus Disease 2019 (COVID-19) vaccine and have no known history of Coronavirus Disease 2019 (COVID-19) or SARS Coronavirus 2 (SARS-CoV-2) infection. They will be assigned to receive COVID-19 vaccine under Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at the 100mcg dose at a 28 days of interval). These pools of participants will be assigned 50 mcg mRNA-1273 at a minimum of 12 weeks following receipt of EUA dosing and followed through 12 months after the last vaccination. A telephone visit will occur one week after each primary EUA vaccination and one week after the booster dose. In person follow-up visits will occur on 14 days following completion of EUA vaccinations and on days 14, and 28 days after the booster dose, as well as 3, 6, and 12 months post the booster vaccination. Additional pools of subjects can be included if needed as additional COVID-19 vaccines are awarded EUA.

New groups may be added to Cohort 1 or 2 dependent upon manufacture of variant lineage spike protein-based vaccine constructs or vaccines newly awarded EUA. The primary objectives of this study are 1) to evaluate the safety and reactogenicity of delayed heterologous or homologous vaccine doses after EUA dosed vaccines, and 2) to evaluate the breadth of the humoral immune responses of heterologous and homologous delayed boost regimens following EUA dosing.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible to participate in this study:

1. Individuals >/= 18 years of age at the time of consent.
2. Received and completed primary mRNA COVID-19 vaccine under EUA dosing guidelines and one or two doses of Ad26.COV2.S at least 12 weeks prior to enrollment (Cohort 1 only).
3. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other study procedures.
4. Determined by medical history, targeted physical examination and clinical judgement of the investigator to be in good health.*

   * Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
5. Female participants of childbearing potential may be enrolled in the study, if all of the following apply:

   * Practiced adequate contraception for 28 days prior to the first dose of vaccine (Day 1),
   * Has agreed to continue adequate contraception through 3 months following the booster dose,
   * Has a negative pregnancy test at screening and on the day of the first study vaccine dose (Day 1),
   * Is not currently breastfeeding.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

1. Known history of SARS-CoV-2 infection. (for Cohort 1 and the primary series of Cohort 2).
2. Prior administration of an investigational coronavirus (SARS Coronavirus (SARS-CoV), Middle East Respiratory Syndrome (MERS-CoV)) vaccine or SARS Coronavirus 2 (SARS-CoV-2) monoclonal antibody in the preceding 90 days or current/planned simultaneous participation in another interventional study.
3. Receipt of SARS Coronavirus 2 (SARS-CoV-2) vaccine prior to study entry (Cohort 2 only).
4. A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine or nanolipid particles.
5. Receipt of any investigational study product within 28 days prior to enrollment.
6. Received or plans to receive a vaccine within 28 days prior to the first dose (Day 1) or plans to receive a non-study vaccine within 28 days prior to or after any dose of study vaccine (with exception for seasonal influenza vaccine within 14 days of study vaccine).
7. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular injections or blood draws, or previously experienced thrombosis with thrombocytopenia (TTS) or heparin-induced thrombocytopenia.
8. Current or previous diagnosis of immunocompromising condition, immune-mediated disease, or other immunosuppressive condition.
9. Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids >/= 20 milligram per day of prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to Day 1.
10. Received immunoglobulin, blood-derived products, within 90 days prior to first study vaccination.
11. An immediate family member or household member of this study's personnel.
12. Is acutely ill or febrile 72 hours prior to or at vaccine dosing (fever defined as >/= 38.0 degrees Celsius or 100.4 degrees Fahrenheit). Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Lyke, M.D., Study Chair — University of Maryland School of Medicine, Center for Vaccine Development and Global Health; Robert L Atmar, M.D., Study Chair — Baylor College of Medicine
Locations (10):
- United States (10):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - University of Maryland Baltimore - Institute of Human Virology, Baltimore, Maryland
  - NYU Langone Vaccine Center, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Atmar RL, Lyke KE, Posavad CM, Deming ME, Brady RC, Dobrzynski D, Edupuganti S, Mulligan MJ, Rupp RE, Rostad CA, Jackson LA, Martin JM, Shriver MC, Rajakumar K, Coler RN, El Sahly HM, Kottkamp AC, Branche AR, Frenck RW, Johnston C, Babu TM, Backer M, Archer JI, Crandon S, Nakamura A, Nayak SU, Szydlo D, Dominguez Islas CP, Brown ER, O'Connell SE, Montefiori DC, Eaton A, Neuzil KM, Stephens DS, Beigel JH, Pasetti M, Roberts PC. Mucosal and Systemic Antibody Responses After Boosting With a Bivalent Messenger RNA Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine. J Infect Dis. 2025 Oct 15;232(4):971-981. doi: 10.1093/infdis/jiaf176. PMID 40298376
- [Derived] Marchese AM, Rousculp M, Macbeth J, Beyhaghi H, Seet BT, Toback S. The Novavax Heterologous Coronavirus Disease 2019 Booster Demonstrates Lower Reactogenicity Than Messenger RNA: A Targeted Review. J Infect Dis. 2024 Aug 16;230(2):e496-e502. doi: 10.1093/infdis/jiad519. PMID 37992183
- [Derived] Lyke KE, Atmar RL, Dominguez Islas C, Posavad CM, Deming ME, Branche AR, Johnston C, El Sahly HM, Edupuganti S, Mulligan MJ, Jackson LA, Rupp RE, Rostad CA, Coler RN, Backer M, Kottkamp AC, Babu TM, Dobrzynski D, Martin JM, Brady RC, Frenck RW Jr, Rajakumar K, Kotloff K, Rouphael N, Szydlo D, PaulChoudhury R, Archer JI, Crandon S, Ingersoll B, Eaton A, Brown ER, McElrath MJ, Neuzil KM, Stephens DS, Post DJ, Lin BC, Serebryannyy L, Beigel JH, Montefiori DC, Roberts PC; DMID 21-0012 Study Group. Immunogenicity of NVX-CoV2373 heterologous boost against SARS-CoV-2 variants. NPJ Vaccines. 2023 Jul 11;8(1):98. doi: 10.1038/s41541-023-00693-z. PMID 37433788
- [Derived] Lyke KE, Atmar RL, Islas CD, Posavad CM, Szydlo D, Paul Chourdhury R, Deming ME, Eaton A, Jackson LA, Branche AR, El Sahly HM, Rostad CA, Martin JM, Johnston C, Rupp RE, Mulligan MJ, Brady RC, Frenck RW Jr, Backer M, Kottkamp AC, Babu TM, Rajakumar K, Edupuganti S, Dobrzynski D, Coler RN, Archer JI, Crandon S, Zemanek JA, Brown ER, Neuzil KM, Stephens DS, Post DJ, Nayak SU, Suthar MS, Roberts PC, Beigel JH, Montefiori DC; DMID 21-0012 Study Group. Rapid decline in vaccine-boosted neutralizing antibodies against SARS-CoV-2 Omicron variant. Cell Rep Med. 2022 Jul 19;3(7):100679. doi: 10.1016/j.xcrm.2022.100679. Epub 2022 Jun 20. PMID 35798000
- [Derived] Atmar RL, Lyke KE, Deming ME, Jackson LA, Branche AR, El Sahly HM, Rostad CA, Martin JM, Johnston C, Rupp RE, Mulligan MJ, Brady RC, Frenck RW Jr, Backer M, Kottkamp AC, Babu TM, Rajakumar K, Edupuganti S, Dobrzynski D, Coler RN, Posavad CM, Archer JI, Crandon S, Nayak SU, Szydlo D, Zemanek JA, Dominguez Islas CP, Brown ER, Suthar MS, McElrath MJ, McDermott AB, O'Connell SE, Montefiori DC, Eaton A, Neuzil KM, Stephens DS, Roberts PC, Beigel JH; DMID 21-0012 Study Group. Homologous and Heterologous Covid-19 Booster Vaccinations. N Engl J Med. 2022 Mar 17;386(11):1046-1057. doi: 10.1056/NEJMoa2116414. Epub 2022 Jan 26. PMID 35081293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants that enrolled in Cohort 1 Group 4E and then rolled over into Cohort 1 Group 15E signed separate informed consent documents prior to successful enrollment in each group. Cohort 1Group 15E referred to as Co 1 Gr 15E below.
Pre-assignment Details: Cohort 1 provided rapid information about the safety, reactogenicity, and immunogenicity of delayed boost in a previously EUA-dosed group. Cohort 2 was an adaptive cohort that was vaccine-naïve that evaluated the safety, reactogenicity and immunogenicity of EUA-dosed vaccine followed by delayed boost.
Groups:
- Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of 100-mcg dose of mRNA-1273 (boost dose). N = 50
  mRNA-1273: 0.5mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose). N = 50
  mRNA-1273: 0.5 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n ˜ 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose). N = 50
  mRNA-1273: 0.5 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp stratified with two age ranges of 18-55 years (n=˜ 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose). N = 50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
- Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2: Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (delayed boost dose). N = 50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
- Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (delayed boost dose). N = 50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
- Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (delayed boost dose). N = 50
  mRNA-1273.211: Lipid nanoparticle (LNP) dispersion containing 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the B.1.351 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273. mRNA-1273.211 (0.2 mg/mL) will be administered in 0.5 mL doses (100 mcg/0.5 mL).
- Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (delayed boost dose). N = 50
  mRNA-1273.211: Lipid nanoparticle (LNP) dispersion containing 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the B.1.351 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273. mRNA-1273.211 (0.2 mg/mL) will be administered in 0.5 mL doses (100 mcg/0.5 mL).
- Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA- 1273 N = 50
  mRNA-1273: 0.25 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  mRNA-1273: 0.25 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  mRNA-1273: 0.25 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp for one or two doses stratified with two age ranges of 18-55 years (n= 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  SARS-CoV-2 rS/M1: SARS-CoV-2 rS Drug Substance containing the prototype Wuhan is formulated with saponin-based Matrix-M adjuvant in a buffer of 25 mM sodium phosphate (pH 7.2), 300 mM sodium chloride, and 0.01% (weight per volume [w/v]) polysorbate 80. NVX-Co-V2373 will be administered in 0.5 mL dose (5 mcg Prototype SARS-CoV-2 rS with 50 mcg Matrix-M adjuvant)
- Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  SARS-CoV-2 rS/M1: SARS-CoV-2 rS Drug Substance containing the prototype Wuhan is formulated with saponin-based Matrix-M adjuvant in a buffer of 25 mM sodium phosphate (pH 7.2), 300 mM sodium chloride, and 0.01% (weight per volume [w/v]) polysorbate 80. NVX-Co-V2373 will be administered in 0.5 mL dose (5 mcg Prototype SARS-CoV-2 rS with 50 mcg Matrix-M adjuvant)
- Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 30) and 56 or older (n = 30) randomized to receive a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2). N =60
  SARS-CoV-2 rS/M1: SARS-CoV-2 rS Drug Substance containing the prototype Wuhan is formulated with saponin-based Matrix-M adjuvant in a buffer of 25 mM sodium phosphate (pH 7.2), 300 mM sodium chloride, and 0.01% (weight per volume [w/v]) polysorbate 80. NVX-Co-V2373 will be administered in 0.5 mL dose (5 mcg Prototype SARS-CoV-2 rS with 50 mcg Matrix-M adjuvant)
- Cohort 2: Prospective cohort with naïve to COVID-19 vaccine and infection participants >/= 18 years of age to receive COVID-19 vaccine intramuscularly under Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at 100mcg dose at 28 day interval) followed by booster vaccination (50 mcg mRNA-1273) after minimum 12 weeks. Second booster administered intramuscular using Moderna mRNA-1273.222 at 50 mcg at 4-12 month interval N=250
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
  mRNA-1273.222: Formulated the same way as the mRNA-1273 vaccine but contains 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273.
Period: All Cohorts Except 15E
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2 | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2
Started | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106
Completed | 50 | 47 | 47 | 31 | 41 | 46 | 48 | 46 | 45 | 35 | 44 | 39 | 43 | 44 | 0 | 10 | 22 | 56
Not Completed | 3 | 4 | 3 | 19 | 8 | 5 | 5 | 5 | 5 | 8 | 6 | 8 | 7 | 2 | 0 | 6 | 9 | 50
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 4 | 1 | 0 | 1 | 2 | 2 | 2 | 4 | 2 | 2 | 0 | 5 | 5 | 28
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 5 | 2 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 1 | 3 | 16
Not completed — Participant relocated, no follow-up planned | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Cohort 1 group 4E Participant rolled over into Cohort 1 group 15E | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant unable to adhere to visit schedule | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Became ineligible after enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Confirmed SARS CoV-2 infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Period: Direct Enroll, Rollover to Co 1 Gr 15E
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2 | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of 100-mcg dose of mRNA-1273 (delayed boost dose). N = 50
  mRNA-1273: 0.5 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (delayed boost dose). N = 50
  mRNA-1273: 0.5 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA) -dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n ˜ 25) randomized to receive a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (delayed boost dose). N = 50
  mRNA-1273: 0.5 mL Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (delayed boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (delayed boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (delayed boost dose). N = 50
  Ad26.COV2.S: Formulated to contain 5x10^10 virus particles of the Ad26 vector encoding the S glycoprotein of SARS-CoV-2. Each dose of the Ad26.COV2.S vaccine also includes sodium chloride, citric acid monohydrate, trisodium citrate dihydrate, polysorbate-80, 2-hydroxypropyl-beta-cyclodextrin, and ethanol. Ad26.COV2.S will be used undiluted to obtain the specified vp content in 0.5 mL doses. Each dose is 0.5 mL.
- Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S 5x10^10 vp stratified with two age ranges of 18-55 years (n=˜ 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (delayed boost dose). N = 50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
- Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna - mRNA-1273 at 100 mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (delayed boost dose). N = 50
  BNT162b2: A nucleoside-modified messenger RNA (modRNA) encoding the viral spike glycoprotein (S) of SARS-CoV-2. Each vial contains up to six doses. BNT162b2 (250 mcg/0.5 mL) will be administered in diluted 0.3 mL doses (30 mcg/0.3 mL).
- Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV.2.S at 5x10^10 vp stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA- 1273 N = 50
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273): Adaptive design cohort with participants that previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30mcg for two doses stratified with two age ranges of 18-55 years (n = 25) and 56 or older (n = 25) randomized to receive a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273. N = 50
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
- Cohort 2: Prospective cohort with naïve to COVID-19 vaccine and infection participants >/= 18 years of age to receive COVID-19 vaccine intramuscularly under Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at 100mcg dose at 28 day interval) followed by delayed booster vaccination (50 mcg mRNA-1273) after minimum 12 weeks. Second booster administered intramuscular using Moderna mRNA-1273.222 at 50 mcg at 4-12 month interval N=250
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike (S) protein of the 2019 novel coronavirus (2019-nCoV).
  mRNA-1273.222: Formulated the same way as the mRNA-1273 vaccine but contains 1:1 mix of mRNAs that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the prefusion stabilized S protein of the Wuhan-Hu-1 strain used in mRNA-1273.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 | Total
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  years
    All Cohorts except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts except 15E | 56.8 (14.5) | 53.1 (16.2) | 54.8 (17.4) | 50.1 (13.9) | 49.9 (16.8) | 50.3 (15.4) | 47.7 (14.5) | 54.3 (16.8) | 50.4 (17.9) | 49.4 (13.6) | 48.3 (16.8) | 48.3 (13.4) | 52.9 (17.2) | 47.8 (16.4) |  | 48.4 (14.7) | 43.2 (11.9) | 39.5 (13.6) | 49.3 (16.0)
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 50.3 (15.9) |  |  |  | 50.3 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  Participants
    All Cohorts Except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts Except 15E: Female | 26 | 32 | 29 | 27 | 16 | 23 | 29 | 26 | 23 | 22 | 23 | 21 | 24 | 27 |  | 6 | 16 | 55 | 425
    All Cohorts Except 15E: Male | 27 | 19 | 21 | 23 | 33 | 28 | 24 | 25 | 27 | 21 | 27 | 26 | 26 | 19 |  | 10 | 15 | 51 | 422
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E: Female |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 9 |  |  |  | 9
    Cohort 1 Group 15E: Male |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 11 |  |  |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  Participants
    All Cohorts Except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts Except 15E: Hispanic or Latino | 4 | 4 | 3 | 2 | 0 | 3 | 2 | 1 | 5 | 1 | 2 | 1 | 2 | 1 |  | 2 | 3 | 5 | 41
    All Cohorts Except 15E: Not Hispanic or Latino | 49 | 46 | 47 | 47 | 49 | 48 | 51 | 50 | 45 | 42 | 47 | 46 | 48 | 45 |  | 14 | 27 | 101 | 802
    All Cohorts Except 15E: Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  | 0 | 1 | 0 | 4
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E: Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2 |  |  |  | 2
    Cohort 1 Group 15E: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 17 |  |  |  | 17
    Cohort 1 Group 15E: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  |  |  | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  Participants
    All Cohorts Except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts Except 15E: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
    All Cohorts Except 15E: Asian | 4 | 5 | 4 | 3 | 5 | 6 | 1 | 2 | 1 | 2 | 6 | 7 | 4 | 7 |  | 0 | 4 | 1 | 62
    All Cohorts Except 15E: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
    All Cohorts Except 15E: Black or African American | 1 | 2 | 3 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 3 | 0 | 4 | 1 |  | 5 | 10 | 32 | 67
    All Cohorts Except 15E: White | 46 | 41 | 43 | 44 | 43 | 40 | 51 | 47 | 43 | 38 | 37 | 40 | 37 | 35 |  | 10 | 15 | 70 | 680
    All Cohorts Except 15E: Multi-Racial | 1 | 3 | 0 | 3 | 1 | 2 | 1 | 0 | 4 | 2 | 3 | 0 | 4 | 3 |  | 1 | 1 | 2 | 31
    All Cohorts Except 15E: Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  | 0 | 1 | 0 | 3
    All Cohorts Except 15E: Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 |  | 0 | 0 | 1 | 4
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 1 Group 15E: Asian |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 1 Group 15E: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 1 Group 15E: Black or African American |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3 |  |  |  | 3
    Cohort 1 Group 15E: White |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 13 |  |  |  | 13
    Cohort 1 Group 15E: Multi-Racial |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4 |  |  |  | 4
    Cohort 1 Group 15E: Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  | 0
    Cohort 1 Group 15E: Other |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  | 0
Height [Mean (Standard Deviation); unit: cm] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  cm
    All Cohorts except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts except 15E | 170.595 (10.875) | 168.104 (10.253) | 169.330 (10.421) | 171.636 (10.273) | 172.547 (9.613) | 170.231 (10.639) | 171.604 (9.582) | 170.448 (9.331) | 171.115 (9.965) | 171.344 (9.844) | 172.266 (10.431) | 173.072 (10.633) | 169.714 (11.691) | 169.990 (8.949) |  | 172.038 (10.676) | 170.835 (10.766) | 171.326 (10.134) | 170.927 (10.203)
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 172.151 (6.268) |  |  |  | 172.151 (6.268)
Weight [Mean (Standard Deviation); unit: kg] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  kg
    All Groups Except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Groups Except 15E | 82.474 (22.586) | 79.960 (17.572) | 82.877 (23.870) | 80.705 (18.437) | 83.536 (20.798) | 80.229 (17.936) | 78.743 (24.710) | 80.766 (17.668) | 80.935 (18.560) | 79.649 (18.894) | 80.050 (19.014) | 81.383 (18.374) | 76.205 (18.407) | 78.521 (18.593) |  | 79.03 (14.60) | 93.17 (26.77) | 88.771 (21.467) | 81.935 (20.458)
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 88.15 (20.08) |  |  |  | 88.15 (20.08)
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: All Cohorts except 15E reported on Row 1, and Cohort 1 Group 15E is reported on Row 2. This is to prevent counting the participants who rolled over into Cohort 1 Group 15E (from Cohort 1 Group 4E) on the same row.
  kg/m2
    All Cohorts except 15E: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 53 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 0 | 16 | 31 | 106 | 847
    All Cohorts except 15E | 28.30 (7.94) | 28.34 (6.10) | 28.79 (7.45) | 27.32 (5.55) | 27.97 (6.40) | 27.58 (5.06) | 26.57 (7.64) | 27.71 (5.21) | 27.76 (6.67) | 26.96 (5.02) | 27.02 (6.61) | 27.01 (4.97) | 26.37 (5.53) | 27.13 (6.08) |  | 26.62 (4.21) | 31.66 (7.73) | 30.36 (7.52) | 27.99 (6.54)
    Cohort 1 Group 15E: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 20
    Cohort 1 Group 15E |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 29.60 (5.84) |  |  |  | 29.60 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Area Under the Curve (AUC) of Antibody Against WA-1 S2-P for Cohort 1
Description: Geometric Mean AUC of Antibody Against WA-1 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method. Units are Electrochemiluminescence (ECL) Signal x 1/dilution (integrated).
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: The mITT population for the population includes all enrolled participants who received the booster vaccine and contributed both pre- and at least one post-vaccination boost venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. When 0 participants are indicated, the assay was not performed for the applicable arm at the time point specified.
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Groups:
- Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of 100-mcg dose of mRNA-1273 (boost dose).
- Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose).
- Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273 (boost dose).
- Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose).
- Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose).
- Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of Ad26.COV2.S 5x10^10 vp (boost dose).
- Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose).
- Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose).
- Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of a 30-mcg dose of BNT162b2 (boost dose).
- Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (boost dose).
- Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of a 100-mcg dose of mRNA-1273.211 (boost dose).
- Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273.
- Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273.
- Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of a 50-mcg dose of mRNA-1273.
- Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Janssen - Ad26.COV2-S 5x10^10 vp, received a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2).
- Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2).
- Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373): Previously (>/=12 weeks) dosed with Emergency Use Authorization (EUA)-dosed vaccination with Pfizer/BioNTech - BNT162b2 at 30 mcg for two doses, received a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2).
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
Arbitrary Unit*1/dilution
  Day 1, Pre-Dose: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
  Day 1, Pre-Dose | 2940.97 [2349.82 to 3680.83] | 26101.97 [22876.53 to 29782.18] | 14223.28 [11259.42 to 17967.32] | 2926.70 [2128.92 to 4023.44] | 20715.09 [17568.48 to 24425.28] | 11549.69 [9316.31 to 14318.48] | 3790.32 [2857.23 to 5028.13] | 23437.84 [20581.58 to 26690.49] | 11448.89 [9385.87 to 13965.38] | 4198.32 [2966.41 to 5941.81] | 12104.83 [9827.34 to 14910.12] | 2314.29 [1712.29 to 3127.94] | 13480.35 [10994.14 to 16528.79] | 8895.46 [7293.62 to 10849.10] | 4423.99 [2495.03 to 7844.25] | 17749.73 [10968.10 to 28724.48] | 13682.64 [8804.30 to 21263.99]
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 22969.71 [15905.34 to 33171.74] | 50130.93 [44100.34 to 56986.18] | 44295.72 [39894.34 to 49182.70]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 46396.64 [43261.81 to 49758.63] | 58170.70 [56455.39 to 59938.12] | 53826.28 [50861.98 to 56963.33] | 11221.56 [9150.39 to 13761.55] | 51277.70 [48148.69 to 54610.04] | 41335.27 [37689.91 to 46688.47] | 42955.92 [39545.96 to 46659.91] | 58564.74 [56547.13 to 60654.33] | 47695.55 [42234.81 to 53862.32] | 49577.25 [45525.67 to 53989.40] | 60745.09 [59183.24 to 62348.16] | 46758.48 [44178.01 to 49489.67] | 59407.62 [57066.79 to 61844.47] | 58728.16 [56832.02 to 60687.56] | 20950.53 [13923.52 to 31523.99] | 46053.86 [38716.71 to 54781.48] | 42857.80 [38031.14 to 48297.02]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 31618.63 [28253.56 to 35384.50] | 47163.57 [44641.79 to 49827.82] | 42511.10 [38846.21 to 46521.74] | 8387.48 [6856.62 to 10260.14] | 49339.52 [45671.10 to 53302.59] | 39977.61 [36170.95 to 44184.88] | 28807.64 [25302.68 to 32798.11] | 48358.86 [45418.40 to 51489.69] | 38564.83 [35140.64 to 42322.68] | 34007.68 [29150.94 to 39673.58] | 48892.87 [45640.19 to 52377.36] | 30620.81 [27303.51 to 34341.16] | 51633.60 [48114.98 to 55409.53] | 47222.88 [43132.31 to 51701.38] | 15093.62 [9651.71 to 23603.84] | 44220.57 [35889.03 to 54486.24] | 38320.95 [30415.62 to 48280.95]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 17458.61 [14702.34 to 20731.61] | 32351.89 [29022.64 to 36063.04] | 28690.99 [24256.45 to 33936.24] | 12896.71 [9184.15 to 18110.00] | 45772.37 [40542.78 to 51676.52] | 35430.22 [30680.95 to 40914.66] | 19889.46 [15887.09 to 24900.12] | 37981.19 [33589.63 to 42946.91] | 28640.42 [24374.56 to 33652.85] | 27894.31 [22343.65 to 34823.87] | 35751.04 [31937.30 to 40020.19] | 20954.21 [17277.95 to 25412.67] | 42109.89 [37225.34 to 47635.38] | 40408.83 [35846.96 to 45551.24] | 20826.02 [12090.96 to 35871.70] | 38984.11 [26907.57 to 56480.79] | 31129.10 [22535.88 to 42999.02]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 24139.14 [16057.25 to 36288.79] | 46337.63 [39831.80 to 53906.06] | 34368.23 [27632.83 to 42745.35] | 20331.28 [14197.27 to 29115.54] | 34556.56 [27979.01 to 42680.42] | 33341.39 [26883.01 to 41351.34] | 25844.56 [19147.02 to 34884.88] | 38808.82 [32552.83 to 46267.09] | 25855.31 [19486.00 to 34306.52] | 45909.39 [40465.43 to 52085.74] | 36651.20 [30142.19 to 44565.78] | 35196.75 [25622.52 to 48348.54] | 43013.25 [30391.43 to 60877.02] | 30573.66 [21592.20 to 43291.02]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 16279.54 [11655.92 to 22737.22] | 30329.85 [23407.80 to 39298.85] | 33164.24 [30222.07 to 49058.36] | 26224.15 [18621.08 to 36931.58] | 47342.92 [41185.51 to 54420.89] | 41154.35 [34353.09 to 49302.13] | 34832.97 [27370.95 to 44329.33] | 37066.79 [30111.92 to 45628.00] | 36487.96 [30305.41 to 43931.79] | 38505.13 [30222.07 to 49058.36] | 46309.04 [39804.39 to 53876.66] | 32151.88 [25389.43 to 40715.52] | 47851.89 [42364.97 to 54049.45] | 44965.48 [38241.12 to 52872.25] | 31119.43 [22820.78 to 42435.85] | 49916.77 [38057.55 to 65471.49] | 37897.76 [26382.63 to 54438.84]

2. Primary Outcome: Geometric Mean of AUC of Antibody Against B.1.351 S2-P for Cohort 1
Description: Geometric Mean AUC of Antibody Against B.1.351 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
Arbitrary Unit*1/dilution
  Day 1, Pre-Dose: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
  Day 1, Pre-Dose | 942.30 [744.40 to 1192.81] | 11013.62 [9254.21 to 13107.54] | 6047.85 [4839.00 to 7558.69] | 954.30 [685.96 to 1327.62] | 8076.74 [6708.27 to 9724.36] | 5201.78 [4221.65 to 6409.48] | 1402.70 [1044.97 to 1882.89] | 10079.24 [8831.54 to 11503.21] | 5572.24 [4706.89 to 6596.69] | 1157.98 [829.29 to 1616.95] | 4842.69 [3832.48 to 6119.18] | 814.66 [600.25 to 1105.67] | 5850.30 [4659.22 to 7345.86] | 4007.33 [3251.91 to 4938.22] | 1525.71 [874.39 to 2662.20] | 8253.24 [4414.58 to 15429.76] | 7414.32 [4422.53 to 12430.01]
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 12221.52 [7549.80 to 19784.06] | 35359.98 [29312.98 to 42654.43] | 29907.22 [25349.53 to 35284.34]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 26285.49 [23490.65 to 29412.84] | 36774.49 [34659.48 to 39018.56] | 34955.90 [32009.83 to 38173.12] | 4374.91 [3521.79 to 5434.68] | 28074.29 [24899.01 to 31654.51] | 21791.31 [18762.06 to 25309.66] | 25833.88 [22966.50 to 29059.26] | 38209.76 [36117.55 to 40423.17] | 30475.16 [26260.31 to 35366.51] | 30963.49 [26929.55 to 35601.69] | 42846.74 [40742.39 to 45059.79] | 26189.91 [23594.30 to 29071.07] | 39348.91 [36296.61 to 42657.88] | 38613.53 [35586.82 to 41897.66] | 10675.96 [6334.38 to 17993.24] | 30089.60 [22836.66 to 39646.08] | 28612.56 [23973.55 to 34149.23]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 15169.94 [13027.23 to 17665.07] | 27671.50 [25424.22 to 30117.43] | 26254.53 [23442.83 to 29403.47] | 2898.58 [2337.97 to 3593.63] | 25421.46 [21951.50 to 29439.92] | 19134.05 [16141.10 to 22681.95] | 14117.54 [12056.77 to 16530.55] | 27268.18 [24809.44 to 29970.60] | 20818.34 [18206.42 to 23804.98] | 19023.81 [15438.33 to 23442.00] | 33082.45 [29822.29 to 36699.02] | 15586.43 [13174.80 to 18439.51] | 33595.91 [30011.95 to 37607.86] | 31546.58 [27868.57 to 35710.00] | 6723.73 [3990.92 to 11327.86] | 26478.42 [19068.38 to 36768.01] | 24620.13 [18379.45 to 32979.82]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 7471.43 [6153.36 to 9071.84] | 15948.35 [13679.33 to 18593.74] | 15594.79 [12707.95 to 19137.42] | 5927.70 [3823.13 to 9190.78] | 25363.92 [20471.42 to 31425.70] | 17961.00 [14221.54 to 22683.74] | 9676.46 [7422.32 to 12615.18] | 20240.62 [17078.35 to 23988.42] | 15227.63 [12263.23 to 18908.62] | 14797.17 [11037.51 to 19837.46] | 21187.80 [18057.84 to 24860.28] | 9654.27 [7577.47 to 12300.25] | 24777.00 [20635.24 to 29750.06] | 24443.88 [20492.73 to 29156.85] | 10607.87 [5511.13 to 20418.12] | 22911.81 [13567.88 to 38690.73] | 19694.67 [13281.97 to 29203.48]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 13419.30 [7963.82 to 22611.94] | 25606.61 [19930.24 to 32899.67] | 18677.11 [13530.91 to 25780.54] | 11200.14 [7325.04 to 17125.25] | 19035.58 [14338.55 to 25271.26] | 19883.25 [15075.44 to 26224.36] | 13779.96 [9225.46 to 20582.97] | 24867.46 [19656.38 to 31460.05] | 13945.30 [9762.02 to 19921.21] | 28289.22 [23181.18 to 34522.83] | 23144.27 [18170.67 to 29479.22] | 20832.94 [13987.12 to 31029.36] | 26049.67 [16237.15 to 41792.13] | 19442.79 [13083.34 to 28893.39]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 8213.69 [5532.02 to 12195.31] | 17151.09 [12218.59 to 24074.79] | 19820.85 [14567.28 to 26969.07] | 14562.44 [9567.57 to 22164.95] | 26463.44 [20623.05 to 33957.80] | 24277.42 [18615.37 to 31661.62] | 21177.37 [15796.85 to 28390.54] | 20937.42 [15870.99 to 27621.20] | 22385.67 [17470.21 to 28684.16] | 23311.90 [17260.46 to 31484.94] | 31525.58 [25510.38 to 38959.13] | 17859.94 [13214.83 to 24137.84] | 30792.74 [25742.82 to 36833.29] | 29301.54 [23585.66 to 36402.65] | 17064.67 [11672.26 to 24948.29] | 31999.19 [21018.85 to 48715.72] | 25344.25 [16274.01 to 39469.76]

3. Primary Outcome: Geometric Mean AUC of Antibody Against B.1.617.2 S2-P for Cohort 1
Description: Geometric Mean AUC of Antibody Against B.1.617.2 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
Arbitrary Unit*1/dilution
  Day 1, Pre-Dose | 1396.82 [1093.87 to 1783.67] | 14461.60 [12217.34 to 17118.11] | 7615.66 [6046.08 to 9592.70] | 1422.80 [1017.63 to 1989.31] | 10772.57 [8973.74 to 12931.97] | 6473.05 [5240.33 to 7995.76] | 1894.19 [1415.79 to 2534.24] | 12682.79 [11027.18 to 14586.97] | 6603.35 [5520.89 to 7898.04] | 1730.28 [1227.75 to 2438.52] | 6229.00 [4948.44 to 7840.96] | 1107.26 [824.30 to 1487.36] | 7371.42 [5895.73 to 9216.47] | 4897.12 [3961.65 to 6053.50] | 2690.71 [1617.54 to 4475.89] | 11890.69 [6800.37 to 20791.30] | 10063.53 [6193.38 to 16352.09]
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 17186.74 [11268.72 to 26212.74] | 41302.86 [35166.31 to 48510.25] | 35909.49 [30979.84 to 41623.57]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 32520.96 [29393.00 to 35981.79] | 42841.53 [40641.10 to 45161.11] | 40054.71 [36657.11 to 43767.22] | 6193.90 [4991.47 to 7685.99] | 35454.71 [32016.76 to 39261.82] | 27283.88 [23749.99 to 31343.58] | 31272.17 [28043.87 to 34872.11] | 43721.86 [41391.13 to 46183.83] | 34878.85 [30128.13 to 40378.68] | 36782.02 [32597.13 to 41504.18] | 48350.60 [46008.19 to 50812.27] | 33526.55 [30717.21 to 36592.83] | 45935.88 [42533.31 to 49610.66] | 45352.29 [42292.27 to 48633.72] | 14825.07 [9202.62 to 23882.64] | 37407.78 [31604.60 to 44276.52] | 34856.19 [29860.57 to 40687.57]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 19450.29 [16870.47 to 22424.61] | 31822.66 [29344.28 to 34510.36] | 29761.16 [26479.16 to 33449.97] | 4208.70 [3415.97 to 5185.39] | 33090.44 [29307.61 to 37361.54] | 24769.12 [21201.21 to 28937.48] | 18843.89 [16118.82 to 22029.67] | 33605.00 [30904.70 to 36541.24] | 26048.76 [23040.07 to 29450.34] | 23195.15 [19169.97 to 28065.51] | 36714.60 [33409.99 to 40346.06] | 19848.42 [17098.69 to 23040.36] | 37238.30 [33422.26 to 41490.05] | 36641.95 [32888.47 to 40823.81] | 9451.28 [5664.54 to 15769.45] | 32383.00 [25355.82 to 41357.72] | 29771.28 [22790.30 to 38890.64]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 10642.97 [8866.09 to 12775.95] | 19755.04 [17184.10 to 22710.63] | 19310.73 [16064.57 to 23212.85] | 8068.78 [5382.52 to 12095.67] | 31914.57 [26757.61 to 38065.43] | 23385.30 [19247.69 to 28412.35] | 12437.92 [9712.65 to 15927.87] | 24536.98 [21093.54 to 28542.55] | 18216.90 [14922.99 to 22237.85] | 19131.14 [14925.42 to 24521.95] | 25309.68 [21792.52 to 29394.49] | 13553.35 [10925.88 to 16812.68] | 29076.21 [24647.52 to 34300.65] | 30020.08 [25781.35 to 34955.70] | 14585.46 [8187.65 to 25982.52] | 28431.40 [18586.62 to 43490.66] | 23753.89 [16497.38 to 34202.24]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 17076.66 [10473.04 to 27844.10] | 32534.84 [26919.75 to 39321.16] | 24178.96 [18403.28 to 31767.28] | 14704.04 [10028.46 to 21559.51] | 23258.35 [18060.99 to 29951.32] | 23893.33 [18564.90 to 30751.12] | 16703.38 [11834.44 to 23575.51] | 28966.27 [23528.68 to 35660.51] | 17723.13 [12813.36 to 24514.19] | 31957.12 [26552.95 to 38461.16] | 27851.85 [22434.81 to 34576.86] | 26576.68 [18819.49 to 37531.31] | 32425.08 [21983.11 to 47826.98] | 24213.35 [16852.99 to 34788.27]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 11447.53 [7975.70 to 16430.64] | 21327.55 [15785.84 to 28814.70] | 24372.65 [18560.59 to 32004.71] | 18956.68 [12843.92 to 27978.66] | 33290.21 [27256.77 to 40659.19] | 30280.41 [24086.36 to 38067.32] | 26161.22 [19977.70 to 34258.68] | 26060.07 [20334.56 to 33397.68] | 27094.44 [21748.26 to 33754.83] | 28150.35 [21687.99 to 36538.30] | 36376.96 [30108.13 to 43951.04] | 22608.60 [17315.37 to 29519.94] | 35405.05 [29961.85 to 41837.12] | 35118.48 [28980.53 to 42556.43] | 21955.78 [15487.15 to 31126.19] | 38608.31 [27513.93 to 54176.26] | 30940.18 [20898.62 to 45806.59]

4. Primary Outcome: Geometric Mean AUC of Antibody Against B.1.1.529 S2-P for Cohort 1
Description: Geometric Mean AUC of Antibody Against B.1.1.529 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
Arbitrary Unit*1/dilution
  Day 1, Pre-Dose: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
  Day 1, Pre-Dose | 355.20 [274.70 to 459.29] | 6123.52 [4971.22 to 7542.92] | 2749.80 [2052.91 to 3683.26] | 350.87 [246.10 to 500.26] | 3749.08 [3022.42 to 4650.45] | 2052.63 [1587.68 to 2653.76] | 502.26 [368.31 to 684.92] | 4295.75 [3567.51 to 5172.65] | 1860.42 [1479.73 to 2339.06] | 484.90 [332.63 to 706.87] | 2128.28 [1648.90 to 2747.05] | 309.27 [227.73 to 420.00] | 2525.90 [1936.94 to 3293.94] | 1579.63 [1248.19 to 1999.08] | 504.21 [254.26 to 999.86] | 3595.20 [1703.38 to 7588.14] | 3106.78 [1690.15 to 5710.79]
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5968.57 [3459.42 to 10297.64] | 21524.83 [15803.89 to 29316.72] | 16656.77 [13114.36 to 21156.05]
  Day 29: number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 17068.46 [14682.35 to 19842.35] | 31782.30 [29363.05 to 34400.87] | 27187.51 [23743.45 to 31131.14] | 1965.71 [1516.28 to 2548.36] | 19054.68 [16009.67 to 22678.84] | 12658.68 [10282.31 to 15584.27] | 16188.16 [13702.59 to 19124.61] | 30886.55 [28161.70 to 33875.05] | 21838.60 [18092.58 to 26360.23] | 22297.06 [18563.04 to 26782.19] | 36401.71 [33873.87 to 39118.19] | 18673.13 [15994.05 to 21800.98] | 34724.95 [31347.16 to 38466.71] | 33890.21 [30923.97 to 37140.98] | 5164.32 [2788.59 to 9564.03] | 17202.81 [11290.70 to 26210.67] | 15484.34 [15484.34 to 20031.40]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 7269.52 [5957.93 to 8869.84] | 18723.69 [16542.78 to 21192.11] | 15312.25 [12688.86 to 18478.02] | 1183.72 [927.65 to 1510.47] | 15698.38 [12689.80 to 19420.25] | 9858.05 [7826.42 to 12417.08] | 7249.59 [5904.49 to 8901.12] | 19202.73 [16618.10 to 22189.36] | 13491.41 [11242.96 to 16189.54] | 9632.54 [7467.24 to 12425.73] | 20953.73 [17953.39 to 24455.47] | 7344.94 [5884.10 to 9168.47] | 22018.09 [18732.94 to 25879.35] | 19275.37 [16140.45 to 23019.18] | 3184.43 [1790.03 to 5665.04] | 14911.93 [8938.59 to 24877.04] | 13089.37 [8831.07 to 19401.00]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 2707.32 [2155.08 to 3401.08] | 7586.78 [6185.95 to 9304.83] | 6807.45 [4485.04 to 9977.37] | 2515.63 [1489.50 to 4248.65] | 12819.14 [9426.83 to 17432.19] | 7831.52 [5710.23 to 10740.85] | 4250.72 [3036.25 to 5950.96] | 11306.69 [8855.84 to 14435.81] | 8133.44 [6106.18 to 10833.76] | 6689.46 [4485.04 to 9977.37] | 10433.04 [8403.37 to 12952.93] | 3979.56 [2902.82 to 5455.69] | 12926.21 [9991.57 to 16722.79] | 12677.50 [9988.16 to 16090.96] | 4536.90 [2151.82 to 9565.60] | 11849.54 [5860.75 to 23957.97] | 9530.78 [5852.57 to 15520.67]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 5675.43 [3026.13 to 10644.13] | 13092.16 [9063.89 to 18910.71] | 8225.58 [5320.59 to 12716.67] | 4637.99 [2773.84 to 7754.96] | 9622.02 [6647.04 to 13928.49] | 10021.44 [6943.97 to 14462.81] | 6073.64 [3512.87 to 10501.12] | 13184.85 [9542.74 to 18217.03] | 5942.40 [3751.38 to 9413.09] | 16035.47 [11998.42 to 21430.86] | 12045.70 [8784.62 to 16517.39] | 9499.76 [5580.83 to 16170.60] | 13423.41 [6703.27 to 26880.61] | 9291.17 [5629.00 to 15335.90]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 3412.16 [2132.56 to 5459.55] | 9039.16 [5869.21 to 13921.20] | 10520.02 [7172.27 to 15430.37] | 6123.72 [3670.11 to 10217.67] | 14026.72 [9872.16 to 19929.68] | 11973.35 [8408.10 to 17050.36] | 9769.74 [6826.15 to 13982.68] | 11132.59 [7711.59 to 16071.22] | 11526.24 [8306.97 to 15993.08] | 11695.26 [7877.62 to 17362.99] | 18446.49 [13727.47 to 24787.74] | 8475.77 [5826.30 to 12330.07] | 17580.65 [13597.51 to 22730.58] | 16727.74 [12527.94 to 22335.47] | 7339.99 [4511.75 to 11941.14] | 17215.73 [9109.88 to 32534.08] | 13220.17 [7525.15 to 23225.18]

5. Primary Outcome: Geometric Mean AUC of Antibody of Antibody Against WA-1 S2-P for Cohort 2
Description: Geometric Mean AUC of Antibody Against WA-1 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: Day 1 Pre-Booster Dose 2, Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: The primary immunogenicity population includes enrolled participants who received all the study vaccines, including the second booster vaccination (Moderna mRNA-1273.222) and who contributed both pre- and at least one post-second booster vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Groups:
- Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222): Naïve to COVID-19 vaccine and infection, received COVID-19 vaccine intramuscularly under Emergency Use Authorization dosing (EUA) (two vaccinations of mRNA-1273 at 100mcg dose at 28 day interval) followed by delayed booster vaccination (50 mcg mRNA-1273) after minimum 12 weeks. Second booster administered intramuscular using Moderna mRNA-1273.222 at 50 mcg at 4-12 month interval
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
Arbitrary Unit*1/dilution
  Day 1, Pre-Booster Vaccination 2 | 193349.76 [136074.53 to 274732.75]
  Day 15: number analyzed (Participants) | 28
  Day 15 | 1201152.28 [899527.72 to 1603915.89]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 921655.60 [684452.31 to 1241063.88]
  Day 91: number analyzed (Participants) | 29
  Day 91 | 688925.53 [520392.79 to 912038.74]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 445271.64 [344427.79 to 575641.23]

6. Primary Outcome: Geometric Mean AUC of Antibody Against BA.1 S2-P for Cohort 2
Description: Geometric Mean AUC of Antibody Against BA.1 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
Arbitrary Unit*1/dilution
  Day 1, Pre-Booster Vaccination 2 | 44367.39 [30868.36 to 63769.67]
  Day 15: number analyzed (Participants) | 28
  Day 15 | 365421.15 [265045.53 to 503810.10]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 260668.10 [185214.52 to 366860.32]
  Day 91: number analyzed (Participants) | 29
  Day 91 | 178509.53 [129548.91 to 245973.92]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 92349.30 [69580.26 to 122569.16]

7. Primary Outcome: Geometric Mean AUC of Antibody Against BA.5 S2-P for Cohort 2
Description: Geometric Mean AUC of Antibody Against BA.5 S2-P using 10-plex ECLIA Assay. Area was computed for electrochemiluminescence signal across sample dilutions using a trapezoidal method.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Unit*1/dilution
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
Arbitrary Unit*1/dilution
  Day 1, Pre-Booster Vaccination 2 | 48314.42 [33707.06 to 69252.05]
  Day 15: number analyzed (Participants) | 28
  Day 15 | 409932.34 [305116.01 to 550756.16]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 297241.68 [219857.75 to 401862.64]
  4Day 91: number analyzed (Participants) | 29
  4Day 91 | 215637.56 [159513.03 to 291509.47]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 128920.81 [98994.66 to 167893.67]

8. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against D614G for Cohort 1
Description: Geometric Mean of Pseudovirus Neutralization against D614G
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
titer
  Day 1, Pre-Dose | 38.68 [26.71 to 56.03] | 378.03 [288.46 to 495.41] | 102.44 [74.23 to 141.38] | 31.27 [20.13 to 48.57] | 254.91 [185.86 to 349.62] | 76.63 [55.25 to 106.28] | 39.01 [26.62 to 57.17] | 238.04 [186.10 to 304.48] | 88.50 [63.17 to 123.98] | 26.82 [16.92 to 42.51] | 66.26 [46.75 to 93.91] | 21.79 [15.82 to 30.00] | 120.75 [85.97 to 169.59] | 55.58 [42.23 to 73.14] | 73.77 [39.67 to 137.16] | 373.44 [140.25 to 994.37] | 342.29 [129.70 to 903.34]
  Day 15: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 49 | 41 | 50 | 43 | 49 | 45 | 19 | 15 | 29
  Day 15 | 2816.89 [2166.33 to 3662.82] | 3758.62 [3043.39 to 4641.93] | 3246.95 [2464.58 to 4277.67] | 129.85 [92.05 to 183.17] | 1578.80 [1200.37 to 2076.54] | 894.14 [652.14 to 1225.94] | 1419.60 [1006.82 to 2001.62] | 2865.92 [2388.29 to 3439.06] | 1806.48 [1379.39 to 2365.81] | 2232.85 [1694.70 to 2941.87] | 3799.17 [2939.29 to 4910.61] | 1804.29 [1444.29 to 2254.03] | 2944.85 [2332.78 to 3717.52] | 2778.25 [2159.32 to 3574.58] | 619.78 [342.68 to 1120.97] | 2431.34 [1407.84 to 4198.95] | 2839.93 [1786.26 to 4515.13]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 49 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 1877.30 [1464.90 to 2405.79] | 2996.19 [2424.66 to 3702.44] | 2138.09 [1624.06 to 2814.81] | 122.76 [92.01 to 163.79] | 2176.45 [1593.18 to 2973.27] | 1090.53 [807.37 to 1472.99] | 1001.61 [784.55 to 1278.72] | 2162.02 [1830.94 to 2552.96] | 1305.46 [1044.34 to 1631.89] | 1686.01 [1271.78 to 2235.15] | 3214.54 [2575.58 to 4012.01] | 1787.22 [1443.66 to 2212.53] | 3383.04 [2673.28 to 4281.24] | 3524.38 [2821.83 to 4401.83] | 499.25 [269.68 to 924.25] | 1978.27 [1024.75 to 3819.03] | 2681.75 [1762.56 to 4080.31]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 816.75 [629.79 to 1059.20] | 1428.84 [1112.25 to 1835.55] | 1142.14 [827.88 to 1575.70] | 120.26 [90.65 to 159.55] | 2659.82 [1943.01 to 3641.09] | 1459.31 [1058.33 to 2012.21] | 598.28 [460.06 to 778.03] | 1179.14 [961.53 to 1446.00] | 845.35 [672.51 to 1062.61] | 689.58 [509.41 to 933.49] | 1308.36 [1002.16 to 1708.11] | 538.84 [417.63 to 695.23] | 1390.28 [1046.31 to 1847.33] | 1208.81 [945.86 to 1544.84] | 305.52 [149.47 to 624.50] | 1661.39 [776.81 to 3553.24] | 1741.71 [949.23 to 3195.82]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 345.65 [256.06 to 466.60] | 599.64 [429.67 to 836.86] | 505.67 [348.87 to 732.94] | 219.40 [124.87 to 385.51] | 1774.79 [1175.90 to 2678.70] | 999.79 [674.16 to 1482.71] | 293.20 [202.20 to 425.14] | 600.34 [450.64 to 799.77] | 476.94 [328.36 to 692.74] | 683.16 [426.84 to 1093.41] | 658.36 [475.86 to 910.84] | 396.82 [281.85 to 558.69] | 962.58 [649.84 to 1425.81] | 1008.89 [707.85 to 1437.94] | 509.25 [208.17 to 1245.80] | 1557.44 [512.62 to 4731.84] | 1356.53 [660.14 to 2787.53]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 36 | 18 | 11 | 22
  Day 273 |  |  |  | 848.73 [400.52 to 1798.52] | 2107.40 [1357.76 to 3270.92] | 1419.20 [822.04 to 2450.16] | 572.36 [292.96 to 1118.21] | 778.99 [475.29 to 1276.74] | 992.82 [619.53 to 1591.02] | 560.75 [290.22 to 1083.43] | 1079.67 [643.56 to 1811.29] | 805.15 [460.85 to 1406.67] | 1475.96 [936.75 to 2325.56] | 1056.44 [651.91 to 1712.00] | 1070.13 [615.88 to 1859.42] | 2340.64 [938.86 to 5835.36] | 1364.44 [686.24 to 2712.92]
  Day 366: number analyzed (Participants) | 49 | 45 | 46 | 30 | 39 | 46 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 407.99 [234.40 to 710.13] | 800.31 [446.29 to 1435.16] | 1006.53 [597.00 to 1696.98] | 807.32 [436.19 to 1494.22] | 2645.09 [1690.99 to 4137.50] | 1982.45 [1267.80 to 3099.95] | 1480.60 [910.31 to 2408.18] | 1341.31 [772.63 to 2328.56] | 1358.34 [840.78 to 2194.47] | 1413.18 [847.65 to 2356.02] | 2068.00 [1235.25 to 3462.14] | 1337.80 [819.28 to 2184.51] | 2597.40 [1541.60 to 4376.28] | 2612.67 [1608.56 to 4243.59] | 650.45 [392.51 to 1077.89] | 2726.20 [1299.43 to 5719.59] | 1532.80 [777.13 to 3023.24]

9. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against B.1.351 for Cohort 1
Description: Geometric Mean of Pseudovirus Neutralization against B.1.351
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: The mITT population for the population includes all enrolled participants who received the booster vaccine and contributed both pre- and at least one post-vaccination boost venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. When 0 participants are indicated, the assay was not performed for the applicable arm at the time point specified. A subset of participants was analyzed for Group 1E-9E and 12E-14E.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 42 | 50 | 20 | 26 | 20 | 19 | 15 | 29
titer
  Day 1, Pre-Dose: number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 42 | 50 | 20 | 20 | 20 | 19 | 15 | 29
  Day 1, Pre-Dose | 8.66 [5.50 to 13.63] | 29.74 [17.80 to 49.69] | 17.81 [13.14 to 24.15] | 6.75 [4.00 to 11.39] | 28.82 [17.22 to 48.23] | 12.06 [7.39 to 19.68] | 7.99 [5.51 to 11.57] | 34.42 [21.87 to 54.17] | 19.67 [12.53 to 30.86] | 8.92 [6.43 to 12.38] | 15.07 [11.29 to 20.11] | 7.76 [5.10 to 11.80] | 41.70 [25.11 to 69.25] | 21.38 [14.17 to 32.24] | 15.60 [8.41 to 28.93] | 77.29 [25.45 to 234.72] | 84.59 [31.88 to 224.50]
  Day 15: number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 41 | 50 | 20 | 26 | 20 | 0 | 0 | 0
  Day 15 | 407.53 [276.66 to 600.31] | 572.08 [358.19 to 913.69] | 582.60 [336.76 to 1007.90] | 24.90 [13.06 to 47.45] | 449.28 [212.80 to 948.58] | 233.11 [130.88 to 415.19] | 332.24 [241.41 to 457.23] | 607.55 [451.31 to 817.89] | 487.02 [340.72 to 696.13] | 362.95 [261.01 to 504.71] | 512.13 [362.77 to 722.99] | 673.88 [415.15 to 1093.86] | 1927.07 [1245.56 to 2981.45] | 1464.22 [870.60 to 2462.60] |  |  |
  Day 29: number analyzed (Participants) | 18 | 20 | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 41 | 50 | 20 | 20 | 19 | 18 | 14 | 29
  Day 29 | 281.66 [188.71 to 420.39] | 439.79 [283.81 to 681.50] | 405.60 [233.58 to 704.32] | 17.61 [10.30 to 30.11] | 394.18 [196.49 to 790.76] | 155.05 [92.99 to 258.54] | 132.44 [103.98 to 168.69] | 398.86 [291.72 to 545.35] | 219.26 [128.70 to 346.61] | 430.23 [305.22 to 606.45] | 899.83 [662.23 to 1222.66] | 275.33 [184.55 to 410.75] | 451.56 [280.55 to 759.36] | 600.49 [343.98 to 1048.27] | 112.57 [52.02 to 243.59] | 568.68 [291.85 to 1108.11] | 1040.55 [631.42 to 1714.78]
  Day 91: number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 19 | 40 | 48 | 19 | 20 | 20 | 19 | 13 | 25
  Day 91 | 117.60 [80.61 to 171.56] | 199.21 [106.69 to 371.97] | 186.12 [106.25 to 326.04] | 13.52 [7.87 to 23.21] | 548.74 [255.67 to 1177.78] | 216.16 [120.84 to 386.66] | 125.92 [78.66 to 201.57] | 252.19 [166.33 to 382.38] | 184.88 [125.71 to 271.92] | 126.92 [91.14 to 176.75] | 343.66 [244.68 to 482.68] | 105.17 [70.33 to 157.26] | 413.72 [223.45 to 766.04] | 223.86 [122.35 to 409.58] | 48.11 [21.96 to 105.44] | 291.20 [116.89 to 725.47] | 408.30 [204.60 to 814.82]
  Day 181: number analyzed (Participants) | 20 | 19 | 19 | 18 | 19 | 20 | 20 | 20 | 16 | 35 | 49 | 20 | 17 | 20 | 0 | 0 | 0
  Day 181 | 46.02 [31.44 to 67.37] | 130.18 [47.43 to 357.26] | 73.97 [40.31 to 125.74] | 54.85 [18.09 to 166.37] | 455.71 [249.68 to 831.76] | 260.07 [134.87 to 501.46] | 68.94 [35.66 to 133.27] | 120.76 [59.11 to 246.73] | 273.59 [96.48 to 775.84] | 174.12 [95.47 to 317.58] | 197.54 [131.19 to 297.45] | 69.40 [34.57 to 139.31] | 327.32 [111.3 to 963.23] | 183.98 [81.95 to 413.02] |  |  |
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 41 | 0 | 0 | 0 | 0 | 0 | 0
  Day 273 |  |  |  |  |  |  |  |  |  | 269.32 [104.3 to 694.56] | 513.05 [265.67 to 990.79] |  |  |  |  |  |
  Day 366: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 44 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366 |  |  |  |  |  |  |  |  |  | 490.51 [267.24 to 900.32] | 856.84 [499.99 to 1631.53] |  |  |  |  |  |

10. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against B.1.617.2 for Cohort 1
Description: Geometric Mean of Pseudovirus Neutralization against B.1.617.2
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: The mITT population for the population includes all enrolled participants who received the booster vaccine and contributed both pre- and at least one post-vaccination boost venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. When 0 participants are indicated, the assay was not performed for the applicable arm at the time point specified. A subset of participants was analyzed for Groups 1E-3E and 10E-11E at Day 29.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 20 | 20 | 46 | 50 | 46 | 0 | 0 | 0
titer
  Day 1, Pre-Dose | 12.02 [8.07 to 17.92] | 101.40 [75.48 to 136.24] | 29.57 [21.58 to 40.50] | 10.27 [6.89 to 15.31] | 107.24 [74.39 to 154.60] | 35.11 [24.73 to 49.83] | 12.63 [8.82 to 18.08] | 90.35 [64.23 to 127.09] | 34.46 [24.32 to 48.84] | 15.00 [8.25 to 27.25] | 48.46 [30.51 to 76.96] | 10.76 [8.53 to 13.57] | 61.98 [41.44 to 92.72] | 23.83 [17.38 to 32.68] |  |  |
  Day 15: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 49 | 0 | 0 | 42 | 48 | 44 | 0 | 0 | 0
  Day 15 | 580.05 [434.90 to 773.64] | 1102.70 [905.86 to 1342.31] | 989.48 [733.87 to 1334.14] | 42.93 [29.64 to 62.17] | 759.42 [565.83 to 1019.25] | 417.81 [290.52 to 600.88] | 490.28 [365.43 to 657.78] | 1525.15 [1239.54 to 1876.57] | 907.09 [676.98 to 1215.41] |  |  | 623.94 [483.45 to 805.25] | 1420.34 [1069.37 to 1886.49] | 1399.37 [1075.48 to 1820.80] |  |  |
  Day 29: number analyzed (Participants) | 20 | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20 | 45 | 46 | 41 | 0 | 0 | 0
  Day 29 | 506.87 [313.85 to 818.59] | 735.02 [507.00 to 1065.60] | 657.82 [384.22 to 1126.28] |  |  |  |  |  |  | 383.22 [246.35 to 596.13] | 1025.81 [698.85 to 1505.75] | 307.44 [249.56 to 378.74] | 782.88 [580.34 to 1056.12] | 781.46 [608.79 to 1003.11] |  |  |

11. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against B.1.1.529 for Cohort 1
Description: Geometric Mean of Pseudovirus Neutralization against B.1.1.529
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 42 | 50 | 46 | 50 | 46 | 19 | 15 | 29
titer
  Day 1, Pre-Dose | 6.04 [5.34 to 6.82] | 28.96 [22.26 to 37.67] | 14.06 [10.50 to 18.82] | 7.18 [5.44 to 9.49] | 20.32 [15.82 to 26.09] | 14.14 [10.59 to 18.88] | 9.01 [6.71 to 12.09] | 23.02 [18.29 to 28.99] | 15.03 [12.29 to 18.38] | 9.20 [6.70 to 12.63] | 15.30 [11.21 to 20.88] | 6.14 [5.27 to 7.14] | 13.94 [10.10 to 19.26] | 10.25 [8.14 to 12.93] | 12.67 [7.09 to 22.66] | 51.38 [15.34 to 172.10] | 84.06 [28.12 to 251.32]
  Day 15: number analyzed (Participants) | 0 | 10 | 0 | 10 | 0 | 10 | 10 | 0 | 10 | 0 | 0 | 0 | 18 | 0 | 19 | 15 | 29
  Day 15 |  | 705.75 [352.82 to 1411.71] |  | 20.23 [9.32 to 43.92] |  | 229.00 [91.27 to 574.57] | 241.39 [123.57 to 471.55] |  | 493.38 [258.09 to 943.16] |  |  |  | 1039.56 [529.84 to 2039.65] |  | 126.81 [61.79 to 260.24] | 749.46 [323.18 to 1738.00] | 816.04 [472.76 to 1408.58]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 240.50 [175.63 to 329.34] | 533.35 [403.74 to 704.57] | 648.16 [440.90 to 952.87] | 26.93 [19.50 to 37.18] | 459.30 [295.56 to 713.75] | 358.92 [249.95 to 515.39] | 238.77 [173.87 to 327.89] | 499.59 [371.65 to 671.57] | 464.12 [341.34 to 631.07] | 395.65 [265.72 to 589.13] | 952.49 [670.44 to 1353.19] | 303.22 [222.61 to 413.02] | 586.83 [425.97 to 808.43] | 1076.92 [784.89 to 1477.59] | 114.81 [51.74 to 254.75] | 704.28 [313.97 to 1579.80] | 1181.12 [639.02 to 2183.10]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 36.18 [26.34 to 49.68] | 100.71 [72.76 to 139.42] | 108.13 [72.31 to 161.69] | 11.15 [8.78 to 14.17] | 180.65 [115.70 to 282.07] | 123.04 [81.81 to 185.02] | 63.64 [46.13 to 87.81] | 183.12 [138.60 to 241.95] | 131.04 [91.52 to 187.61] | 136.63 [91.99 to 202.91] | 368.11 [256.47 to 528.36] | 89.71 [62.51 to 128.74] | 247.05 [170.31 to 358.38] | 406.30 [286.71 to 575.77] | 82.90 [38.02 to 180.79] | 589.29 [248.62 to 1396.74] | 627.30 [307.69 to 1278.94]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 31.78 [23.21 to 43.52] | 73.17 [49.15 to 108.95] | 72.58 [47.71 to 110.42] | 76.78 [40.61 to 145.14] | 499.15 [295.81 to 842.26] | 339.84 [194.48 to 593.83] | 80.65 [50.79 to 128.05] | 140.61 [87.05 to 227.13] | 170.76 [100.43 to 290.34] | 217.99 [109.36 to 434.51] | 222.76 [136.84 to 362.65] | 66.61 [38.45 to 115.38] | 175.75 [97.08 to 318.14] | 307.56 [170.82 to 553.77] | 209.59 [69.70 to 630.27] | 360.07 [63.89 to 2029.20] | 753.27 [299.16 to 1896.69]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 36 | 18 | 11 | 22
  Day 273 |  |  |  | 223.89 [90.67 to 552.84] | 480.51 [240.17 to 961.35] | 364.66 [181.21 to 733.83] | 157.27 [73.05 to 338.59] | 159.41 [86.09 to 295.18] | 324.05 [177.60 to 591.24] | 150.67 [59.57 to 381.09] | 254.41 [121.74 to 531.66] | 258.14 [118.81 to 560.88] | 421.76 [215.93 to 823.79] | 333.17 [173.11 to 641.21] | 859.98 [386.11 to 1915.39] | 1221.74 [418.03 to 3570.65] | 1012.61 [456.88 to 2244.31]
  Day 366: number analyzed (Participants) | 49 | 45 | 46 | 30 | 39 | 46 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 102.18 [53.54 to 194.99] | 232.18 [107.17 to 503.01] | 353.35 [183.42 to 680.70] | 203.18 [98.77 to 417.96] | 483.16 [261.67 to 892.13] | 566.71 [295.77 to 1085.87] | 575.70 [311.61 to 1063.60] | 239.69 [119.72 to 479.88] | 442.53 [242.01 to 809.19] | 835.72 [433.04 to 1612.89] | 1048.01 [502.09 to 2187.54] | 518.33 [258.81 to 1038.08] | 725.75 [381.49 to 1380.67] | 1052.87 [565.12 to 1961.59] | 648.36 [407.78 to 1030.88] | 1307.88 [652.45 to 2621.71] | 1201.30 [545.41 to 2645.94]

12. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against D614G for Cohort 2
Description: Geometric Mean of Pseudovirus Neutralization against D614G
Time Frame: Day 1 Pre-Vaccination 1, Day 43 Post-Vaccination 1, Day 15 Post-Booster Dose 1, Day 1 Pre-Booster Dose 2, Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
titer
  Day 1, Pre-Vaccination 1 | 13.23 [6.82 to 25.67]
  Day 43, Post Vaccination 1 | 4010.57 [2785.54 to 5774.35]
  Day 15, Post Booster Vaccination 1 | 7456.62 [4647.00 to 11964.94]
  Day 1, Pre-Booster Vaccination 2 | 2225.56 [1468.38 to 3373.20]
  Day 15, Post-Booster Vaccination 2: number analyzed (Participants) | 28
  Day 15, Post-Booster Vaccination 2 | 18927.45 [13150.29 to 27242.60]
  Day 29, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 29, Post-Booster Vaccination 2 | 17481.83 [11657.50 to 26216.11]
  Day 91, Post-Booster Vaccination 2: number analyzed (Participants) | 29
  Day 91, Post-Booster Vaccination 2 | 9244.35 [6596.46 to 12955.15]
  Day 181, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 181, Post-Booster Vaccination 2 | 3932.11 [2993.93 to 5164.27]

13. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against BA.1 for Cohort 2
Description: Geometric Mean of Pseudovirus Neutralization against BA.1
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
titer
  Day 1, Pre-Vaccination 1 | 6.36 [4.51 to 8.96]
  Day 43, Post Vaccination 1 | 189.09 [100.15 to 357.04]
  Day 15, Post Booster Vaccination 1 | 2680.27 [1368.13 to 5250.85]
  Day 1, Pre-Booster Vaccination 2 | 679.09 [376.79 to 1223.91]
  Day 15, Post-Booster Vaccination 2: number analyzed (Participants) | 28
  Day 15, Post-Booster Vaccination 2 | 12381.92 [7615.21 to 20132.34]
  Day 29, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 29, Post-Booster Vaccination 2 | 9496.08 [5113.33 to 17635.40]
  Day 91, Post-Booster Vaccination 2: number analyzed (Participants) | 29
  Day 91, Post-Booster Vaccination 2 | 3272.98 [2290.23 to 4677.44]
  Day 181, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 181, Post-Booster Vaccination 2 | 4076.50 [2337.99 to 7107.76]

14. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against BA.4/5 for Cohort 2
Description: Geometric Mean of Pseudovirus Neutralization against BA.4/5
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
titer
  Day 1, Pre-Vaccination 1 | 7.59 [4.83 to 11.93]
  Day 43, Post Vaccination 1 | 260.47 [141.07 to 480.92]
  Day 15, Post Booster Vaccination 1 | 1377.38 [854.38 to 2220.54]
  Day 1, Pre-Booster Vaccination 2 | 464.55 [253.81 to 850.28]
  Day 15, Post-Booster Vaccination 2: number analyzed (Participants) | 28
  Day 15, Post-Booster Vaccination 2 | 10328.08 [6854.83 to 15561.19]
  Day 29, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 29, Post-Booster Vaccination 2 | 7558.08 [4947.10 to 11547.08]
  Day 91, Post-Booster Vaccination 2: number analyzed (Participants) | 29
  Day 91, Post-Booster Vaccination 2 | 6848.36 [4320.84 to 10854.38]
  Day 181, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 181, Post-Booster Vaccination 2 | 2540.36 [1707.64 to 3779.15]

15. Primary Outcome: Geometric Mean of Pseudovirus Neutralization Against XBB.1 for Cohort 2
Description: Geometric Mean of Pseudovirus Neutralization against XBB.1
Time Frame: as for outcome 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
titer
  Day 1, Pre-Vaccination 1 | 5.28 [4.72 to 5.91]
  Day 43, Post Vaccination 1 | 24.37 [14.01 to 42.37]
  Day 15, Post Booster Vaccination 1 | 132.74 [75.92 to 232.10]
  Day 1, Pre-Booster Vaccination 2 | 39.52 [24.28 to 64.33]
  Day 15, Post-Booster Vaccination 2: number analyzed (Participants) | 28
  Day 15, Post-Booster Vaccination 2 | 969.29 [576.68 to 1629.20]
  Day 29, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 29, Post-Booster Vaccination 2 | 648.84 [389.17 to 1081.76]
  Day 91, Post-Booster Vaccination 2: number analyzed (Participants) | 29
  Day 91, Post-Booster Vaccination 2 | 462.50 [288.10 to 742.47]
  Day 181, Post-Booster Vaccination 2: number analyzed (Participants) | 27
  Day 181, Post-Booster Vaccination 2 | 211.99 [135.32 to 332.10]

16. Primary Outcome: Frequency of Any Unsolicited Adverse Events (AEs)
Description: Number of participants who experienced any unsolicited AEs through 28 days post vaccination
Time Frame: Day 1 through Day 29 for Cohort 1, 28 days post any vaccination in Cohort 2
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 28 | 29 | 31 | 31 | 28 | 28 | 28 | 29 | 24 | 22 | 24 | 20 | 30 | 25 | 8 | 6 | 14 | 60

17. Primary Outcome: Frequency of Any Protocol Specified Adverse Events of Special Interest (AESIs)
Description: Number of participants that experienced any AESIs during the course of the study. An adverse event of special interest (serious or nonserious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor is required. AESIs include anosmia, ageusia, subacute thyroiditis, acute pancreatitis, appendicitis, rhabdomyolysis, acute respiratory distress syndrome, coagulation disorders, acute cardiovascular injury, acute kidney injury, acute liver injury, dermatologic findings, multisystem inflammatory disorders, thrombocytopenia, acute aseptic arthritis, new onset of or worsening of neurologic disease, anaphylaxis, and other syndromes.
Time Frame: For Cohort 1, Day 1 through Day 366; for Cohort 2, Day 1 through Day 590
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 5

18. Primary Outcome: Frequency of Any New-onset Chronic Medical Conditions (NOCMCs)
Description: Number of participants that experienced any NOCMCs during the course of the study
Time Frame: For Cohort 1, Day 1 through Day 366; for Cohort 2, Day 1 through Day 590
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 0 | 6 | 2 | 3 | 3 | 1 | 1 | 4 | 2 | 2 | 0 | 2 | 3 | 1 | 0 | 0 | 2 | 2

19. Primary Outcome: Number of Participants With Any Medically-attended Adverse Events (MAAEs)
Description: Number of participants that experienced MAAEs during the course of the study.
Time Frame: For Cohort 1, Day 1 through Day 366; for Cohort 2, Day 1 through Day 590
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

20. Primary Outcome: Frequency of Any Serious Adverse Events (SAEs)
Description: The number of participants that experience any SAEs from Day 1 to study completion. An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in: death, a lifethreatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: For Cohort 1, Day 1 through Day 366; for Cohort 2, Day 1 through Day 590
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 2 | 4 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 5

21. Primary Outcome: Frequency of Systemic Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any systemic solicited AEs through 7 days post any vaccination. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever.
Time Frame: Day 1 through Day 8 for Cohort 1, and through 7 days post any vaccination for Cohort 2
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 38 | 47 | 45 | 39 | 42 | 42 | 39 | 38 | 46 | 37 | 38 | 41 | 42 | 40 | 17 | 10 | 23 | 93

22. Primary Outcome: Frequency of Local Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any local solicited AEs through 7 days post any vaccination. Local events include: pain at injection site, erythema, and induration.
Time Frame: Day 1 through Day 8 for Cohort 1, and through 7 days post any vaccination for Cohort 2
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Group 16E (Boost mRNA-1273, Boost NVX-CoV2373): Previously (>/=12 weeks) received Emergency Use Authorization (EUA)-dosed vaccination with Moderna-mRNA-1273 at 100mcg for two doses, received a single intramuscular (IM) injection of a 5-mcg dose of NVX-CoV2373 (SARS-COV-2).
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Boost mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 43 | 50 | 47 | 50 | 46 | 20 | 16 | 31 | 106
Participants | 41 | 44 | 41 | 38 | 35 | 35 | 48 | 39 | 45 | 39 | 45 | 42 | 41 | 40 | 11 | 5 | 16 | 94

23. Primary Outcome: Percent of Participants Who Seroconverted Against WA-1 S2-P for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against WA-1 S2-P
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 58 [33 to 80] | 47 [21 to 73] | 45 [26 to 64]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 94 [84 to 99] | 12 [4 to 24] | 37 [23 to 52] | 46 [31 to 61] | 15 [6 to 28] | 45 [31 to 60] | 88 [77 to 96] | 14 [6 to 26] | 50 [36 to 64] | 90 [77 to 97] | 68 [53 to 80] | 100 [92 to 100] | 55 [40 to 69] | 80 [65 to 90] | 44 [22 to 69] | 43 [18 to 71] | 45 [26 to 64]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 50 | 51 | 51 | 47 | 40 | 48 | 42 | 49 | 46 | 19 | 13 | 25
  Day 91 | 88 [76 to 96] | 6 [1 to 17] | 26 [15 to 40] | 25 [14 to 40] | 15 [6 to 28] | 43 [31 to 60] | 78 [65 to 89] | 8 [2 to 19] | 26 [14 to 40] | 83 [67 to 93] | 46 [31 to 61] | 86 [71 to 95] | 48 [34 to 63] | 59 [43 to 73] | 32 [13 to 57] | 38 [14 to 68] | 40 [21 to 61]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 65 [51 to 78] | 2 [1 to 11] | 8 [2 to 20] | 50 [35 to 65] | 9 [2 to 21] | 40 [26 to 55] | 60 [44 to 74] | 6 [1 to 17] | 22 [11 to 36] | 60 [42 to 76] | 31 [18 to 45] | 82 [68 to 92] | 36 [22 to 52] | 52 [37 to 67] | 47 [24 to 71] | 27 [6 to 61] | 26 [10 to 48]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 84 [64 to 95] | 14 [5 to 30] | 38 [22 to 55] | 51 [34 to 68] | 10 [3 to 24] | 31 [17 to 48] | 46 [28 to 66] | 34 [20 to 51] | 88 [72 to 97] | 50 [32 to 68] | 57 [39 to 73] | 61 [36 to 83] | 36 [11 to 69] | 27 [11 to 50]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 56 [41 to 70] | 7 [1 to 18] | 26 [14 to 41] | 83 [65 to 94] | 18 [8 to 34] | 47 [32 to 62] | 78 [64 to 89] | 11 [4 to 25] | 35 [21 to 51] | 75 [57 to 89] | 52 [37 to 68] | 85 [69 to 94] | 44 [28 to 60] | 70 [54 to 83] | 67 [41 to 87] | 50 [19 to 81] | 35 [15 to 59]

24. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.351 S2-P for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against B.1.351 S2-P
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 50 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 84 [60 to 97] | 53 [27 to 79] | 55 [36 to 74]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 98 [90 to 99] | 33 [21 to 48] | 76 [61 to 87] | 56 [41 to 71] | 35 [22 to 51] | 47 [33 to 62] | 96 [87 to 99] | 43 [29 to 58] | 72 [58 to 84] | 98 [87 to 99] | 90 [78 to 97] | 100 [92 to 100] | 78 [63 to 88] | 87 [73 to 95] | 78 [52 to 94] | 50 [23 to 77] | 52 [33 to 71]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 50 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 94 [84 to 99] | 16 [7 to 29] | 50 [36 to 94] | 35 [22 to 51] | 34 [21 to 49] | 43 [29 to 58] | 84 [71 to 93] | 25 [14 to 40] | 38 [25 to 54] | 95 [83 to 99] | 76 [65 to 90] | 98 [87 to 99] | 68 [53 to 80] | 83 [69 to 92] | 42 [20 to 67] | 46 [19 to 75] | 48 [28 to 69]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 75 [61 to 86] | 4 [1 to 14] | 16 [7 to 30] | 50 [35 to 65] | 44 [30 to 60] | 48 [34 to 63] | 74 [60 to 86] | 12 [5 to 24] | 26 [14 to 41] | 80 [63 to 92] | 51 [36 to 66] | 87 [73 to 95] | 43 [28 to 59] | 63 [48 to 77] | 63 [38 to 84] | 36 [11 to 39] | 30 [13 to 53]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 80 [59 to 93] | 46 [29 to 63] | 54 [37 to 71] | 65 [47 to 80] | 26 [13 to 42] | 46 [30 to 63] | 68 [48 to 84] | 59 [42 to 74] | 94 [80 to 99] | 68 [49 to 83] | 68 [50 to 82] | 72 [47 to 90] | 45 [17 to 77] | 36 [17 to 59]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 68 [53 to 80] | 20 [10 to 35] | 48 [33 to 63] | 87 [69 to 96] | 49 [32 to 65] | 53 [38 to 68] | 85 [71 to 94] | 25 [13 to 40] | 60 [44 to 75] | 94 [79 to 99] | 70 [55 to 83] | 92 [79 to 98] | 68 [52 to 82] | 79 [64 to 90] | 78 [52 to 94] | 60 [26 to 88] | 50 [27 to 73]

25. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.617.2 S2-P for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against B.1.617.2 S2-P
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 50 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 68 [43 to 87] | 53 [27 to 79] | 52 [33 to 71]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 96 [87 to 99] | 27 [16 to 42] | 67 [52 to 80] | 48 [33 to 63] | 27 [15 to 42] | 51 [37 to 65] | 96 [87 to 99] | 39 [26 to 54] | 70 [55 to 82] | 95 [83 to 99] | 88 [76 to 95] | 100 [92 to 100] | 71 [57 to 83] | 87 [73 to 95] | 61 [36 to 83] | 50 [23 to 77] | 48 [29 to 67]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 50 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 90 [79 to 97] | 6 [1 to 17] | 40 [26 to 55] | 31 [19 to 46] | 26 [14 to 40] | 51 [37 to 65] | 86 [74 to 94] | 22 [11 to 35] | 38 [25 to 54] | 93 [80 to 98] | 77 [63 to 88] | 98 [87 to 99] | 66 [51 to 79] | 74 [59 to 86] | 32 [13 to 57] | 46 [19 to 75] | 36 [18 to 57]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 73 [59 to 84] | 2 [1 to 11] | 18 [9 to 32] | 50 [35 to 65] | 31 [18 to 47] | 50 [36 to 64] | 64 [49 to 77] | 12 [5 to 24] | 28 [16 to 43] | 83 [66 to 93] | 49 [34 to 64] | 91 [79 to 98] | 41 [26 to 57] | 61 [45 to 75] | 58 [33 to 80] | 36 [11 to 69] | 30 [13 to 53]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 80 [59 to 93] | 37 [21 to 55] | 51 [34 to 68] | 62 [45 to 78] | 23 [11 to 39] | 46 [30 to 63] | 68 [48 to 84] | 56 [40 to 72] | 94 [80 to 99] | 65 [46 to 80] | 65 [47 to 80] | 72 [47 to 90] | 45 [17 to 77] | 27 [11 to 50]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 68 [53 to 80] | 18 [8 to 32] | 46 [31 to 61] | 87 [69 to 96] | 38 [23 to 55] | 58 [42 to 72] | 85 [71 to 94] | 25 [13 to 40] | 60 [44 to 75] | 88 [71 to 96] | 70 [55 to 83] | 92 [79 to 98] | 66 [49 to 80] | 77 [61 to 88] | 72 [47 to 90] | 60 [26 to 88] | 40 [19 to 64]

26. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.1.529 S2-P for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against B.1.1.529 S2-P
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 50 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 15 | 29
  Day 15 |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 84 [60 to 97] | 60 [32 to 84] | 59 [39 to 76]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 50 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 100 [93 to 100] | 63 [48 to 76] | 92 [80 to 98] | 69 [54 to 81] | 63 [47 to 76] | 57 [42 to 71] | 98 [90 to 99] | 78 [65 to 89] | 96 [86 to 99] | 98 [87 to 99] | 96 [86 to 99] | 100 [92 to 100] | 92 [80 to 98] | 98 [88 to 99] | 86 [65 to 99] | 50 [23 to 77] | 52 [33 to 71]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 50 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 90 [79 to 97] | 28 [16 to 42] | 68 [53 to 80] | 38 [24 to 53] | 53 [38 to 68] | 55 [40 to 69] | 94 [84 to 99] | 49 [35 to 63] | 79 [64 to 89] | 95 [83 to 99] | 85 [72 to 94] | 98 [87 to 99] | 78 [64 to 88] | 91 [79 to 98] | 68 [43 to 87] | 46 [19 to 75] | 52 [31 to 72]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 75 [61 to 86] | 6 [1 to 17] | 20 [10 to 34] | 50 [35 to 65] | 47 [32 to 62] | 48 [34 to 63] | 70 [55 to 83] | 28 [16 to 42] | 52 [37 to 67] | 77 [60 to 90] | 59 [44 to 73] | 82 [68 to 92] | 57 [41 to 72] | 72 [57 to 84] | 63 [38 to 84] | 36 [11 to 69] | 30 [13 to 53]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 37 | 18 | 11 | 22
  Day 273 |  |  |  | 84 [64 to 95] | 63 [45 to 79] | 54 [37 to 71] | 57 [39 to 73] | 38 [23 to 55] | 56 [40 to 72] | 68 [48 to 84] | 66 [49 to 80] | 91 [76 to 98] | 68 [49 to 83] | 73 [56 to 86] | 78 [52 to 94] | 45 [17 to 77] | 36 [17 to 59]
  Day 366: number analyzed (Participants) | 50 | 45 | 46 | 30 | 39 | 45 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 66 [51 to 79] | 31 [18 to 47] | 54 [39 to 69] | 87 [66 to 96] | 62 [45 to 77] | 62 [49 to 76] | 85 [71 to 94] | 48 [32 to 63] | 60 [44 to 75] | 97 [84 to 99] | 70 [55 to 83] | 92 [79 to 98] | 73 [57 to 86] | 81 [67 to 92] | 78 [52 to 94] | 60 [26 to 88] | 50 [27 to 73]

27. Primary Outcome: Percent of Participants Who Seroconverted Against WA-1 S2-P for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against WA-1 S2-P
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15: number analyzed (Participants) | 28
  Day 15 | 61 [41 to 78]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 56 [35 to 75]
  Day 91 | 41 [24 to 61]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 26 [11 to 46]

28. Primary Outcome: Percent of Participants Who Seroconverted Against BA.1 S2-P for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against BA.1 S2-P
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15: number analyzed (Participants) | 28
  Day 15 | 79 [59 to 92]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 70 [50 to 86]
  Day 91 | 38 [21 to 58]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 19 [6 to 38]

29. Primary Outcome: Percent of Participants Who Seroconverted Against BA.5 S2-P for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against BA.5 S2-P
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15: number analyzed (Participants) | 28
  Day 15 | 79 [59 to 92]
  Day 29: number analyzed (Participants) | 27
  Day 29 | 70 [50 to 86]
  Day 91 | 45 [26 to 64]
  Day 181: number analyzed (Participants) | 27
  Day 181 | 37 [19 to 58]

30. Primary Outcome: Percent of Participants Who Seroconverted Against D614G for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against D614G
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 50 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 49 | 41 | 50 | 43 | 49 | 45 | 19 | 15 | 29
  Day 15 | 100 [93 to 100] | 84 [71 to 93] | 100 [93 to 100] | 50 [36 to 64] | 61 [46 to 75] | 82 [69 to 91] | 98 [90 to 99] | 94 [84 to 99] | 98 [89 to 99] | 98 [87 to 99] | 100 [93 to 100] | 100 [92 to 100] | 98 [89 to 99] | 100 [92 to 100] | 63 [43 to 87] | 67 [38 to 88] | 55 [36 to 74]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 49 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 94 [84 to 99] | 80 [67 to 90] | 100 [93 to 100] | 54 [39 to 69] | 73 [59 to 85] | 80 [67 to 90] | 94 [84 to 99] | 90 [79 to 97] | 90 [78 to 97] | 98 [87 to 99] | 98 [89 to 99] | 100 [92 to 100] | 98 [89 to 99] | 100 [92 to 100] | 72 [47 to 90] | 50 [23 to 77] | 55 [36 to 74]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 90 [79 to 97] | 42 [28 to 57] | 86 [73 to 94] | 44 [29 to 59] | 74 [60 to 86] | 88 [76 to 96] | 84 [71 to 93] | 57 [42 to 71] | 72 [57 to 84] | 95 [83 to 99] | 90 [77 to 97] | 95 [84 to 99] | 84 [71 to 93] | 98 [88 to 99] | 53 [29 to 76] | 46 [19 to 75] | 52 [31 to 72]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 73 [59 to 84] | 14 [6 to 27] | 49 [34 to 64] | 57 [41 to 72] | 64 [49 to 78] | 78 [64 to 88] | 62 [46 to 75] | 28 [16 to 42] | 57 [41 to 71] | 83 [66 to 93] | 78 [63 to 88] | 91 [79 to 98] | 66 [50 to 80] | 87 [74 to 95] | 58 [33 to 80] | 36 [11 to 69] | 52 [31 to 73]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 36 | 18 | 11 | 22
  Day 273 |  |  |  | 72 [51 to 88] | 63 [45 to 79] | 73 [56 to 86] | 62 [45 to 78] | 51 [35 to 68] | 64 [47 to 79] | 75 [55 to 89] | 73 [57 to 86] | 94 [80 to 99] | 76 [59 to 89] | 83 [67 to 94] | 78 [52 to 94] | 45 [17 to 77] | 41 [21 to 64]
  Day 366: number analyzed (Participants) | 49 | 45 | 46 | 30 | 39 | 46 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 57 [42 to 71] | 38 [24 to 53] | 57 [41 to 71] | 80 [61 to 92] | 69 [52 to 83] | 83 [69 to 92] | 85 [71 to 94] | 61 [45 to 76] | 77 [61 to 88] | 88 [71 to 96] | 84 [70 to 93] | 95 [83 to 99] | 85 [71 to 94] | 93 [81 to 99] | 72 [47 to 90] | 60 [26 to 88] | 50 [27 to 73]

31. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.351 for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against B.1.351
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 41 | 50 | 20 | 20 | 20 | 19 | 14 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 41 | 50 | 20 | 20 | 20 | 0 | 0 | 0
  Day 15 | 95 [75 to 99] | 95 [75 to 99] | 100 [83 to 100] | 40 [19 to 64] | 90 [68 to 99] | 100 [83 to 100] | 100 [83 to 100] | 95 [75 to 99] | 95 [75 to 99] | 98 [87 to 99] | 98 [89 to 99] | 100 [83 to 100] | 100 [83 to 100] | 100 [83 to 100] |  |  |
  Day 29: number analyzed (Participants) | 18 | 20 | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 41 | 50 | 20 | 20 | 19 | 18 | 14 | 29
  Day 29 | 94 [73 to 99] | 95 [75 to 99] | 100 [82 to 100] | 40 [19 to 64] | 80 [56 to 94] | 95 [75 to 99] | 95 [75 to 99] | 85 [62 to 97] | 95 [75 to 99] | 100 [91 to 100] | 100 [93 to 100] | 100 [83 to 100] | 85 [62 to 97] | 100 [82 to 100] | 61 [36 to 83] | 64 [35 to 87] | 59 [39 to 76]
  Day 91: number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 19 | 40 | 48 | 19 | 20 | 20 | 19 | 13 | 25
  Day 91 | 85 [62 to 97] | 80 [56 to 94] | 95 [75 to 99] | 20 [6 to 44] | 80 [56 to 94] | 95 [75 to 99] | 90 [68 to 99] | 70 [46 to 88] | 79 [54 to 94] | 95 [83 to 99] | 94 [83 to 99] | 89 [67 to 99] | 80 [56 to 94] | 80 [56 to 94] | 47 [24 to 71] | 46 [19 to 75] | 52 [31 to 72]
  Day 181: number analyzed (Participants) | 20 | 19 | 19 | 18 | 19 | 20 | 20 | 20 | 16 | 35 | 49 | 20 | 17 | 20 | 0 | 0 | 0
  Day 181 | 65 [41 to 85] | 32 [13 to 57] | 53 [29 to 76] | 56 [31 to 78] | 79 [54 to 94] | 90 [68 to 99] | 65 [41 to 85] | 35 [15 to 59] | 69 [41 to 89] | 77 [60 to 90] | 82 [68 to 91] | 75 [51 to 91] | 59 [33 to 82] | 65 [41 to 85] |  |  |
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 41 | 0 | 0 | 0 | 0 | 0 | 0
  Day 273 |  |  |  |  |  |  |  |  |  | 79 [59 to 92] | 83 [68 to 93] |  |  |  |  |  |
  Day 366: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 44 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366 |  |  |  |  |  |  |  |  |  | 91 [75 to 98] | 93 [81 to 99] |  |  |  |  |  |

32. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.617.2 for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against B.1.617.2
Time Frame: Day 15, Day 29
Population: The mITT population for the population includes all enrolled participants who received the booster vaccine and contributed both pre- and at least one post-vaccination boost venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. When 0 participants are indicated, the assay was not performed for the applicable arm at the time point specified. This assay was not completed for Group 15E, 16E, and 17E.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273)
Number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 49 | 20 | 20 | 45 | 48 | 44
percentage of participants
  Day 15: number analyzed (Participants) | 53 | 51 | 50 | 50 | 49 | 50 | 52 | 51 | 49 | 0 | 0 | 42 | 48 | 44
  Day 15 | 94 [84 to 99] | 86 [74 to 94] | 100 [93 to 100] | 56 [41 to 70] | 65 [50 to 78] | 74 [60 to 85] | 96 [87 to 99] | 88 [76 to 96] | 94 [83 to 99] |  |  | 100 [92 to 100] | 92 [80 to 98] | 100 [92 to 100]
  Day 29: number analyzed (Participants) | 20 | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20 | 45 | 46 | 41
  Day 29 | 90 [68 to 99] | 70 [46 to 88] | 100 [83 to 100] |  |  |  |  |  |  | 90 [68 to 99] | 100 [83 to 100] | 98 [88 to 99] | 83 [69 to 92] | 100 [91 to 100]

33. Primary Outcome: Percent of Participants Who Seroconverted Against B.1.1.529 for Cohort 1
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against B.1.1.529
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 273, Day 366
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373)
Number analyzed (Participants) | 52 | 51 | 50 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 50 | 46 | 19 | 15 | 29
percentage of participants
  Day 15: number analyzed (Participants) | 0 | 10 | 0 | 10 | 0 | 10 | 10 | 0 | 10 | 0 | 0 | 0 | 18 | 0 | 19 | 15 | 29
  Day 15 |  | 90 [55 to 99] |  | 40 [12 to 74] |  | 100 [69 to 100] | 100 [69 to 100] |  | 100 [48 to 100] |  |  |  | 94 [73 to 99] |  | 79 [54 to 94] | 87 [60 to 98] | 55 [36 to 74]
  Day 29: number analyzed (Participants) | 52 | 51 | 49 | 48 | 48 | 51 | 52 | 51 | 50 | 41 | 50 | 46 | 49 | 45 | 18 | 14 | 29
  Day 29 | 100 [93 to 100] | 92 [81 to 98] | 98 [89 to 99] | 52 [37 to 67] | 92 [80 to 98] | 98 [90 to 99] | 92 [81 to 98] | 94 [84 to 99] | 98 [89 to 99] | 95 [83 to 99] | 98 [89 to 99] | 100 [92 to 100] | 98 [89 to 99] | 100 [92 to 100] | 83 [59 to 96] | 86 [57 to 98] | 66 [46 to 82]
  Day 91: number analyzed (Participants) | 51 | 50 | 50 | 48 | 47 | 51 | 51 | 51 | 47 | 40 | 48 | 42 | 50 | 46 | 19 | 13 | 25
  Day 91 | 67 [52 to 79] | 46 [32 to 61] | 72 [58 to 84] | 17 [7 to 30] | 68 [53 to 93] | 76 [63 to 87] | 76 [63 to 87] | 80 [67 to 90] | 74 [60 to 86] | 90 [76 to 97] | 92 [80 to 98] | 93 [81 to 99] | 92 [81 to 98] | 96 [85 to 99] | 74 [49 to 91] | 69 [39 to 91] | 56 [35 to 76]
  Day 181: number analyzed (Participants) | 52 | 49 | 49 | 44 | 45 | 50 | 47 | 50 | 46 | 35 | 49 | 45 | 44 | 46 | 19 | 11 | 23
  Day 181 | 56 [41 to 70] | 31 [18 to 45] | 59 [44 to 73] | 61 [45 to 76] | 82 [68 to 92] | 88 [76 to 95] | 68 [53 to 81] | 52 [37 to 66] | 74 [59 to 86] | 83 [66 to 93] | 78 [63 to 88] | 67 [51 to 80] | 66 [50 to 80] | 93 [82 to 99] | 68 [43 to 87] | 55 [23 to 83] | 57 [34 to 77]
  Day 273: number analyzed (Participants) | 0 | 0 | 0 | 25 | 35 | 37 | 37 | 39 | 39 | 28 | 41 | 33 | 34 | 36 | 18 | 11 | 22
  Day 273 |  |  |  | 76 [55 to 91] | 83 [66 to 93] | 70 [53 to 84] | 62 [45 to 78] | 51 [35 to 68] | 82 [66 to 92] | 61 [41 to 78] | 66 [49 to 80] | 85 [68 to 95] | 85 [69 to 95] | 89 [74 to 97] | 94 [73 to 99] | 82 [48 to 98] | 64 [41 to 83]
  Day 366: number analyzed (Participants) | 49 | 45 | 46 | 30 | 39 | 46 | 46 | 44 | 43 | 32 | 44 | 39 | 41 | 43 | 18 | 10 | 20
  Day 366 | 65 [50 to 78] | 51 [36 to 66] | 78 [64 to 89] | 80 [61 to 92] | 77 [61 to 89] | 83 [69 to 92] | 89 [76 to 96] | 66 [50 to 80] | 79 [64 to 90] | 97 [84 to 99] | 89 [75 to 96] | 85 [69 to 94] | 88 [74 to 96] | 93 [81 to 99] | 89 [65 to 99] | 70 [35 to 93] | 55 [32 to 77]

34. Primary Outcome: Percent of Participants Who Seroconverted Against D614G for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Dose 1 against D614G
Time Frame: Day 43 Post-Dose 1, Day 15 Post Booster Dose 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
percentage of participants
  Day 43 Post-Dose 1 | 97 [83 to 99]
  Day 15 Post Booster Dose 1 | 100 [88 to 100]

35. Primary Outcome: Percent of Participants Who Seroconverted Against BA.1 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Dose 1 against BA.1
Time Frame: Day 43 Post-Dose 1, Day 15 Post Booster Dose 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
percentage of participants
  Day 43 Post-Dose 1 | 97 [83 to 99]
  Day 15 Post Booster Dose 1 | 100 [88 to 100]

36. Primary Outcome: Percent of Participants Who Seroconverted Against BA.4/5 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Dose 1 against BA.4/5
Time Frame: Day 43 Post-Dose 1, Day 15 Post Booster Dose 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
percentage of participants
  Day 43 Post-Dose 1 | 97 [83 to 99]
  Day 15 Post Booster Dose 1 | 87 [83 to 99]

37. Primary Outcome: Percent of Participants Who Seroconverted Against XBB.1 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Dose 1 against XBB.1
Time Frame: Day 43 Post-Dose 1, Day 15 Post Booster Dose 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 30
percentage of participants
  Day 43 Post-Dose 1 | 47 [28 to 66]
  Day 15 Post Booster Dose 1 | 93 [78 to 99]

38. Primary Outcome: Percent of Participants Who Seroconverted Against D614G for Cohort 2
Description: as for outcome 34
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15 Post-Booster Dose 2: number analyzed (Participants) | 28
  Day 15 Post-Booster Dose 2 | 71 [51 to 87]
  Day 29 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 29 Post-Booster Dose 2 | 74 [54 to 89]
  Day 91 Post-Booster Dose 2 | 45 [26 to 64]
  Day 181 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 181 Post-Booster Dose 2 | 22 [9 to 42]

39. Primary Outcome: Percent of Participants Who Seroconverted Against BA.1 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Booster Dose 2 against BA.1
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15 Post-Booster Dose 2: number analyzed (Participants) | 28
  Day 15 Post-Booster Dose 2 | 86 [67 to 96]
  Day 29 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 29 Post-Booster Dose 2 | 89 [71 to 98]
  Day 91 Post-Booster Dose 2 | 59 [39 to 76]
  Day 181 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 181 Post-Booster Dose 2 | 59 [39 to 78]

40. Primary Outcome: Percent of Participants Who Seroconverted Against BA.4/5 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Booster Dose 2 against BA.4/5
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15 Post-Booster Dose 2: number analyzed (Participants) | 28
  Day 15 Post-Booster Dose 2 | 89 [72 to 98]
  Day 29 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 29 Post-Booster Dose 2 | 89 [71 to 98]
  Day 91 Post-Booster Dose 2 | 90 [73 to 98]
  Day 181 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 181 Post-Booster Dose 2 | 48 [29 to 68]

41. Primary Outcome: Percent of Participants Who Seroconverted Against XBB.1 for Cohort 2
Description: Percent of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from Pre-Booster Dose 2 against XBB.1
Time Frame: Day 15 Post-Booster Dose 2, Day 29 Post-Booster Dose 2, Day 91 Post-Booster Dose 2, Day 181 Post-Booster Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (Vaccine naïve, Received Moderna mRNA-1273.222)
Number analyzed (Participants) | 29
percentage of participants
  Day 15 Post-Booster Dose 2: number analyzed (Participants) | 28
  Day 15 Post-Booster Dose 2 | 93 [76 to 99]
  Day 29 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 29 Post-Booster Dose 2 | 93 [76 to 99]
  Day 91 Post-Booster Dose 2 | 79 [69 to 92]
  Day 181 Post-Booster Dose 2: number analyzed (Participants) | 27
  Day 181 Post-Booster Dose 2 | 48 [29 to 68]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from the time of each vaccination through 7 days post each vaccination. Participants were also assessed for delayed onset local reactions through 14 days post each vaccination. Unsolicited AEs of all severities were reported from the time of study product administration through 28 days post each vaccination. SAEs, AESIs, MAAEs and NOCMCs were reported from the time of study product administration through end of study (Day 366 for Cohort 1 and Day 590 for Cohort 2).
Description: After 28 days post last vaccination through the end of planned study participation, only SAEs, AESIs, MAAEs, and NOCMCs will be reported as AEs; end of planned study participation for Cohort 1 is Day 366 and for Cohort 2 is Day 590. For the 12 participants that rolled over from Cohort 1 Group 4E into Cohort 1 Group 15E, any adverse events that were reported are counted based on the group that they were enrolled in at the time of the event.
Arm/Group | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/51 | 0/50 | 0/50 | 0/49 | 0/51 | 0/52 | 0/51 | 0/50 | 0/43 | 0/50 | 0/47 | 0/50 | 0/46 | 0/20 | 0/16 | 0/31 | 0/106
Serious Adverse Events (participants affected / at risk) | 2/53 | 4/51 | 0/50 | 1/50 | 1/49 | 2/51 | 1/52 | 1/51 | 0/50 | 0/43 | 2/50 | 1/47 | 1/50 | 1/56 | 0/20 | 0/16 | 1/31 | 5/106
Other Adverse Events (participants affected / at risk) | 49/53 | 49/51 | 50/50 | 46/50 | 46/49 | 47/51 | 52/52 | 50/51 | 50/50 | 43/43 | 48/50 | 46/47 | 49/50 | 46/46 | 18/20 | 12/16 | 27/31 | 100/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) (N=53) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) (N=51) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) (N=50) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) (N=50) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) (N=49) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) (N=51) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) (N=52) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) (N=51) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) (N=50) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) (N=43) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) (N=50) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) (N=47) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) (N=50) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) (N=56) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) (N=20) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) (N=16) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) (N=31) | Cohort 2 (N=106)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Group 1E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273) (N=53) | Cohort 1 Group 2E (Prime mRNA-1273, Boost 100 mcg mRNA-1273) (N=51) | Cohort 1 Group 3E (Prime BNT162b2, Boost 100 mcg mRNA-1273) (N=50) | Cohort 1 Group 4E (Prime Ad26.COV2.S, Boost Ad26.COV2.S) (N=50) | Cohort 1 Group 5E (Prime mRNA-1273, Boost Ad26.COV2.S) (N=49) | Cohort 1 Group 6E (Prime BNT162b2, Boost Ad26.COV2.S) (N=51) | Cohort 1 Group 7E (Prime Ad26.COV2.S, Boost BNT162b2) (N=52) | Cohort 1 Group 8E (Prime mRNA-1273, Boost BNT162b2) (N=51) | Cohort 1 Group 9E (Prime BNT162b2, Boost BNT162b2) (N=50) | Cohort 1 Group 10E (Prime Ad26.COV2.S, Boost 100 mcg mRNA-1273.211) (N=43) | Cohort 1 Group 11E (Prime BNT162b2, Boost 100 mcg mRNA-1273.211) (N=50) | Cohort 1 Group 12E (Prime Ad26.COV2.S, Boost 50 mcg mRNA-1273) (N=47) | Cohort 1 Group 13E (Prime mRNA-1273, Boost 50 mcg mRNA-1273) (N=50) | Cohort 1 Group 14E (Prime BNT162b2, Boost 50 mcg mRNA-1273) (N=46) | Cohort 1 Group 15E (Prime Ad26.COV2.S, Boost NVX-CoV2373) (N=20) | Cohort 1 Group 16E (Prime mRNA-1273, Boost NVX-CoV2373) (N=16) | Cohort 1 Group 17E (Prime BNT162b2, Boost NVX-CoV2373) (N=31) | Cohort 2 (N=106)
Nausea (Gastrointestinal disorders) | 9 (9) | 10 (10) | 11 (11) | 9 (9) | 12 (12) | 9 (9) | 7 (7) | 8 (8) | 7 (7) | 7 (7) | 12 (12) | 7 (7) | 11 (11) | 6 (6) | 5 (5) | 4 (4) | 1 (1) | 43 (55)
Chills (General disorders) | 11 (11) | 22 (22) | 23 (23) | 9 (9) | 23 (23) | 16 (16) | 8 (8) | 3 (3) | 10 (10) | 12 (12) | 24 (24) | 6 (6) | 15 (15) | 20 (20) | 2 (2) | 2 (2) | 4 (4) | 66 (98)
Injection site induration (General disorders) | 8 (16) | 9 (18) | 5 (10) | 2 (4) | 0 (0) | 4 (7) | 3 (6) | 7 (14) | 2 (3) | 1 (2) | 4 (8) | 3 (5) | 2 (4) | 5 (10) | 1 (2) | 0 (0) | 0 (0) | 19 (50)
Injection site pain (General disorders) | 41 (41) | 44 (44) | 41 (41) | 38 (38) | 35 (35) | 35 (35) | 48 (48) | 37 (37) | 45 (45) | 39 (39) | 45 (45) | 42 (42) | 41 (41) | 40 (40) | 11 (11) | 5 (5) | 15 (15) | 93 (220)
Malaise (General disorders) | 35 (35) | 40 (40) | 37 (37) | 31 (31) | 38 (38) | 38 (38) | 35 (35) | 34 (34) | 40 (40) | 34 (34) | 36 (36) | 31 (31) | 36 (36) | 33 (33) | 13 (13) | 7 (7) | 13 (13) | 80 (172)
Pyrexia (General disorders) | 5 (10) | 8 (16) | 12 (24) | 2 (4) | 15 (30) | 11 (22) | 2 (4) | 1 (2) | 4 (8) | 4 (8) | 15 (30) | 1 (2) | 6 (12) | 9 (18) | 0 (0) | 0 (0) | 0 (0) | 21 (52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 19 (19) | 18 (18) | 11 (11) | 16 (16) | 20 (20) | 7 (7) | 9 (9) | 10 (10) | 13 (13) | 16 (16) | 7 (7) | 13 (13) | 11 (11) | 3 (3) | 3 (3) | 4 (4) | 53 (81)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 38 (38) | 35 (35) | 25 (25) | 32 (32) | 31 (31) | 22 (22) | 22 (22) | 26 (26) | 27 (27) | 27 (27) | 25 (25) | 30 (30) | 29 (29) | 8 (8) | 4 (4) | 16 (16) | 78 (145)
Headache (Nervous system disorders) | 16 (16) | 33 (33) | 32 (32) | 25 (25) | 26 (26) | 23 (23) | 18 (18) | 28 (28) | 24 (24) | 18 (18) | 27 (27) | 20 (20) | 21 (21) | 24 (24) | 10 (10) | 3 (3) | 6 (6) | 73 (123)
Injection site erythema (General disorders) | 2 (4) | 6 (12) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 2 (4) | 2 (4) | 1 (2) | 1 (2) | 5 (10) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 2 (4) | 12 (27)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 2 (4)
Bradycardia (Cardiac disorders) | 5 (5) | 4 (5) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 4 (6) | 2 (2) | 2 (2) | 4 (6) | 1 (1) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 4 (5) | 4 (4) | 4 (4) | 3 (4) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 6 (6)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Blood pressure systolic increased (Investigations) | 3 (3) | 6 (6) | 2 (2) | 5 (6) | 4 (4) | 2 (2) | 5 (7) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 15 (18)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Systolic hypertension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Micrognathia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (5) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT04889209/Prot_003.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT04889209/SAP_002.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04889209/ICF_001.pdf